CLINICAL TRIAL: NCT02409342
Title: A Phase III, Open Label, Randomized Study of Atezolizumab (Anti-PD-L1 Antibody) Compared With a Platinum Agent (Cisplatin or Carboplatin) in Combination With Either Pemetrexed or Gemcitabine for PD-L1-Selected, Chemotherapy-Naive Patients With Stage IV Non-Squamous Or Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of Atezolizumab (MPDL3280A) Compared With a Platinum Agent (Cisplatin or Carboplatin) + (Pemetrexed or Gemcitabine) in Participants With Stage IV Non-Squamous or Squamous Non-Small Cell Lung Cancer (NSCLC) [IMpower110]
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29431; 2014-003083-21 (EudraCT Number)
Record Dates: First submitted 2015-04-01; First posted 2015-04-06 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer, Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — atezolizumab; Carboplatin; Cisplatin; Gemcitabine; Pemetrexed

ARMS (2):
- (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) (Active Comparator): Participants with non-squamous NSCLC will receive chemotherapy with pemetrexed in combination with either cisplatin or carboplatin (per investigator discretion) on Day 1 of each 21-day cycle for 4 or 6 cycles as per local standard of care, followed by maintenance therapy with pemetrexed alone as per local standard of care until disease progression (per RECIST v1.1), unacceptable toxicity, or death (maximum up to approximately 58 months). Participants with squamous NSCLC will receive chemotherapy with gemcitabine on Days 1 and 8 of each 21-day cycle in combination with either cisplatin or carboplatin on Day 1 of each 21-day cycle for 4 or 6 cycles as per local standard of care, followed by best supportive care as per local standard of care until disease progression, unacceptable toxicity, or death (maximum up to approximately 58 months).
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Gemcitabine; Drug: Pemetrexed
- Atezolizumab (Experimental): Participants with squamous or non-squamous NSCLC will receive atezolizumab on Day 1 of each 21-day cycle until loss of clinical benefit (as assessed by the investigator), unacceptable toxicity, or death (maximum up to approximately 58 months).
  Interventions: Drug: Atezolizumab (MPDL3280A) [TECENTRIQ], an engineered anti-PDL1 antibody

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A) [TECENTRIQ], an engineered anti-PDL1 antibody — Atezolizumab 1200 milligram (mg) will be administered as intravenous infusion every 21 days until loss of clinical benefit (as assessed by the investigator), unacceptable toxicity, or death (maximum up to approximately 58 months).
  Other Names: MPDL3280A, RO5541267
  Arms: Atezolizumab
Drug: Carboplatin — Carboplatin will be administered as intravenous infusion at a dose of area under the concentration-time curve (AUC) 6 when given in combination with pemetrexed or at a dose of AUC 5 when given in combination with gemcitabine, every 21 days for 4 or 6 cycles as per local standard of care.
  Arms: (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine)
Drug: Cisplatin — Cisplatin will be administered as intravenous infusion at a dose of 75 mg per meter squared (mg/m^2) every 21 days for 4 or 6 cycles as per local standard of care.
  Arms: (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine)
Drug: Gemcitabine — Gemcitabine will be administered as intravenous infusion at a dose of 1250 mg/m^2 (in combination with cisplatin) or 1000 mg/m^2 (in combination with carboplatin), on Days 1 and 8 of each 21-day cycle for 4 or 6 cycles as per local standard of care.
  Arms: (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine)
Drug: Pemetrexed — Pemetrexed will be administered as intravenous infusion at a dose of 500 mg/m^2 on Day 1 of each 21-day cycle as per local standard of care until disease progression (per RECIST v1.1), unacceptable toxicity, or death (maximum up to approximately 58 months).
  Arms: (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine)

SUMMARY:
This randomized, open-label study will evaluate the efficacy and safety of atezolizumab compared with chemotherapy consisting of a platinum agent (cisplatin or carboplatin per investigator discretion) combined with either pemetrexed (non-squamous disease) or gemcitabine (squamous disease) in programmed death-ligand 1 (PD-L1)-selected, chemotherapy-naive participants with Stage IV Non-Squamous or Squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, Stage IV non-squamous or squamous NSCLC
* No prior treatment for Stage IV non-squamous or squamous NSCLC. Participant known to have a sensitizing mutation in the epidermal growth factor receptor (EGFR) gene or an anaplastic lymphoma kinase (ALK) fusion oncogene are excluded from the study
* Tumor PD-L1 expression as determined by immunohistochemistry (IHC) assay of archival tumor tissue or tissue obtained at screening
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
* Adequate hematologic and end-organ function

Exclusion Criteria:

* Known sensitizing mutation in the EGFR gene or ALK fusion oncogene
* Active or untreated central nervous system (CNS) metastases as determined by Computed Tomography (CT) or magnetic resonance imaging (MRI) evaluation
* Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome
* Pregnant or lactating women
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Positive test for Human Immunodeficiency Virus (HIV)
* Active hepatitis B or hepatitis C
* Prior treatment with cluster of differentiation (CD) 137 agonists or immune checkpoint blockade therapies, anti PD1, and anti-PD-L1 therapeutic antibody
* Severe infection within 4 weeks prior to randomization
* Significant history of cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2022-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (142):
- United States (9):
  - University of California San Diego, La Jolla, California
  - Yale Cancer Center, New Haven, Connecticut
  - Lynn Cancer Institute - West, Boca Raton, Florida
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Oregon Health & Science Uni, Portland, Oregon
  - Sarah Cannon Cancer Center, Germantown, Tennessee
  - Vanderbilt University Medical Center; Multiple Sclerosis Center, Nashville, Tennessee
  - Hematology Oncology Associates of Fredericksburg, Inc., Fredericksburg, Virginia
  - VA Puget Sound Health Care Sys, Seattle, Washington
- Brazil (11):
  - Centro de Pesquisas Clinicas em Oncologia - CPCO, Cachoeiro de Itapemirim, Espírito Santo
  - Oncovida*X, Salvador, Estado de Bahia
  - Instituto Nacional de Cancer - INCa; Oncologia, Rio de Janeiro, Rio de Janeiro
  - Associacao Hospital de Caridade Ijui*X; Departamento De Oncologia, Ijuí, Rio Grande do Sul
  - Hospital da Cidade de Passo Fundo; Centro de Pesquisa em Oncologia, Passo Fundo, Rio Grande do Sul
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Instituto Joinvilense de Hematologia E Oncologia, Joinville, Santa Catarina
  - *X*Fundacao PIO XII, Barretos, São Paulo
  - Instituto Do Câncer Do Estado de São Paulo Octávio Frias de Oliveira, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo
- Harbin Medical University Tumor Hospital, Harbin, China
- France (10):
  - CHU Angers, Angers
  - Hospital d Instructions des Armees Percy, Clamart
  - Hôpital Universitaire Dupuytren, Limoges
  - Clinique Clémentville, Montpellier
  - Centre D'oncologie de Gentilly, Nancy
  - Hopital Tenon, Paris
  - Centre Hospitalier Regional La Reunion Site Felix Guyon, Saint-Denis
  - Hopital d'Instruction des Armees de Begin, Saint-Mandé
  - Centre Hospitalier Regional Sud Reunion, Saint-Pierre
  - Centre Paul Strauss, Strasbourg
- Germany (2):
  - Asklepios-Fachklinik Muenchen-Gauting; Klinik Für Pneumologie, Gauting
  - Pius-Hospital Oldenburg, Oldenburg
- Greece (11):
  - Sotiria Chest Hospital of Athens, Athens
  - IASO General Hospital of Athens, Athens
  - Metropolitan Hospital, Athens
  - Attikon University General Hospital, Chaïdári
  - University General Hospital of Larissa, Larissa
  - University General Hospital of Patras, Pátrai
  - Thermi Clinic, Thermi, Thessaloniki
  - Bioclinic Thessaloniki, Thessaloniki
  - EUROMEDICA General Clinic of Thessaloniki; Gastroenterology Department, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
  - Georgios Papanikolaou General Hosp. of Thessaloniki, Thessaloniki
- Hungary (4):
  - Uzsoki Utcai Korhaz, Budapest
  - Szabolcs-Szatmar-Bereg Megyei; Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Pecsi Tudomanyegyetem, Pécs
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet; Megyei Onkologiai Kozpont, Szolnok
- Italy (12):
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Centro Di Riferimento Oncologico; Struttura Operativa Complessa Di Oncologia Medica B, Aviano, Friuli Venezia Giulia
  - Asst Papa Giovanni XXIII, Bergamo, Lombardy
  - Azienda Ospedaliera Istituti Ospitalieri, Cremona, Lombardy
  - Ospedale San Raffaele S.r.l., Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale ? ASST di Monza, Monza, Lombardy
  - Istituto Nazionale dei Tumori, Monza, Lombardy
  - Istituto Clinico Humanitas, Rozzano (MI), Lombardy
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Azienda Ospedaliero-Universitaria ?PoliclinicoVittorio Emanuele?- P.O. G. Rodolico; Oncologia Medica, Catania, Sicily
  - Azienda Ospedaliera Universitaria Integrata Verona; UOC Oncologia, Verona, Veneto
- Japan (16):
  - Aichi Cancer Center Hospital; Respiratory Medicine, Aichi
  - Nagoya University Hospital; Respiratory Medicine, Aichi
  - Kyushu University Hospital; Respiratory, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - Kobe City Medical Center General Hospital; Respiratory Medicine, Hyōgo
  - Hyogo Cancer Center; Thoracic Oncology, Hyōgo
  - Ibaraki Prefectural Central Hospital; Division of respiratory, Ibaraki
  - Sendai Kousei Hospital; Pulmonary Medicine, Miyagi
  - Okayama University Hospital; Respiratory and Allergy Medicine, Okayama
  - Osaka International Cancer Institute; Thoracic Oncology, Osaka
  - Kansai Medical university Hospital; Thoracic Oncology, Osaka
  - Osaka Habikino Medical Center, Osaka
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakaishi
  - Saitama Cancer Center; Thoracic Oncology, Satima
  - National Cancer Center Hospital; Thoracic Medical Oncology, Tokyo
  - Tokyo Medical University Hospital; Dept of Surgery, Tokyo
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Warminsko-Mazurskie Centrum Chorób P?uc w Olsztynie; Oddzial onkologii z pododdzialem chemioterapii, Olsztyn
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii w Poznaniu, Poznan
  - Med-Polonia Sp. z o.o., Poznan
- Romania (7):
  - Teo Health SA - Saint Constantin Hospital, Brasov
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
  - Oncology Center Sf. Nectarie, Craiova
  - Institutul Regional de Oncologie Iasi; Clinica de Hematologie, Iași
  - Sibiu Emergency Clinical County Hospital, Sibiu
  - Oncocenter Clinical Oncology, Timi?oara
  - Oncomed SRL, Timișoara
- Russia (11):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk, Arhangelsk
  - Federal State Institution Medical Radiology Research Center, Obninsk, Kaluga Oblast
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Principal Military Clinical Hospital n.a. N.N. Burdenko, Moscow, Moscow Oblast
  - Saint Petersburg Clinical Hospital of the Russian Academy of Sciences, Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Ministry of Healthcare of Tatarstan Republic, Kazan', Tatarstan Republic
  - Regional Clinical Oncology Center, Ryazan
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - St. Petersburg Med Univ; n.a. I.P. Pavlov; Pulmonology Research, Saint Petersburg
  - Mordovia State University, Saransk
  - Volgograd Regional Clinical Oncology Dispensary, Volgograd
- Serbia (4):
  - Clinical Center of Serbia, Belgrade
  - Institute for Oncology and Radiology of Serbia; Medical Oncology, Belgrade
  - Institute of Lung Diseases Vojvodina, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
- South Korea (3):
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kangbuk Samsung Hospital, Seoul
- Spain (15):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Consorcio Hospitalario Provincial de Castellon, Castellon de LA Plana/castello de LA Plana, Castellon
  - Hospital Universitario A Coruña, A Coruña, LA Coruña
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Clinico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hosp Clinico Univ Lozano Blesa; División De Oncología Médica, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- Thailand (4):
  - Prince of Songkla University; Department Of Internal Medicine, Faculty Of Medicine, Hat Yai
  - Khon Kaen University, Khon Kaen
  - Chiang Rai Prachanukroh Hospital, Muang
  - Buddhachinnaraj Hospital, Phitsanulok
- Turkey (Türkiye) (6):
  - Cukurova University Medical Faculty Balcali Hospital, Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Izmir Dr. Suat Seren Gogus Hastaliklari ve Cerrahisi Egitim ve Arastirma Hastanesi, Izmir
  - Inonu University Faculty of Medicine Turgut Ozal Medical Center, Malatya
- Ukraine (8):
  - Municipal Noncommercial Institution Regional Center of Oncology, Kharkiv, Kharkiv Governorate
  - Municipal Noncomercial Enterprise Odessa Regional Oncology Center ofthe Odessa StateAdministration, Odesa, Kherson Governorate
  - Municipal non profit enterprise of Sumy Regional Council Sumy Regional Clinical Oncology Disp, Sumy, Kholm Governorate
  - Communal Non-profit Enterprise City Clinical Hospital #4 of Dnipro City Council - PPDS; Chemotherapy, Dnipro, KIEV Governorate
  - Kyiv Railway Clinical Hospital #3 of Branch Health Center of the PJSC Ukrainian Railway, Kyiv, KIEV Governorate
  - Communal Nonprofit Enterprise Podilsky Regional Center Of Oncology OfTheVinnytsia Regional Council, Vinnytsia, KIEV Governorate
  - The Municipal Enterprise Volyn Regional Medical Oncology Centre of the Volyn Regional Council, Lutsk, Volhynian Governorate
  - Private Enterprise Private Manufacturing Company Acinus, Kirovograd
- United Kingdom (3):
  - Birmingham Heartlands Hospital, Birmingham
  - Colchester General Hospital, Colchester, Essex
  - Christie Hospital, Manchester

REFERENCES:
- [Derived] Li B, Rong D, Lin H. Atezolizumab monotherapy as first-line treatment for non-small cell lung cancer ineligible for treatment with a platinum-containing regimen (IPSOS): a cost-effectiveness analysis in the USA. BMJ Open. 2024 Nov 12;14(11):e083716. doi: 10.1136/bmjopen-2023-083716. PMID 39532375
- [Derived] Herbst RS, Giaccone G, de Marinis F, Reinmuth N, Vergnenegre A, Barrios CH, Morise M, Felip E, Andric Z, Geater S, Ozguroglu M, Zou W, Sandler A, Enquist I, Komatsubara K, Deng Y, Kuriki H, Wen X, McCleland M, Mocci S, Jassem J, Spigel DR. Atezolizumab for First-Line Treatment of PD-L1-Selected Patients with NSCLC. N Engl J Med. 2020 Oct 1;383(14):1328-1339. doi: 10.1056/NEJMoa1917346. PMID 32997907

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment included: Japan (16 centers), Spain (15 centers), Greece (12 centers), Italy (12 centers), Brazil (11 centers), Russian (11 centers), France (10 centers), United States of America (9 centers), Ukraine (8 centers), Romania (7 centers), Turkey (6 centers), Poland (5 centers), Serbia (5 centers), Hungary (4 centers), Thailand (4 centers), Great Britain (3 centers), Republic of Korea (3 centers), Germany (2 centers), China (1 center).
Pre-assignment Details: Study is considered 'Completed' because all of the criteria for End of Study have been met. Participants in survival follow-up completed their last visit and participants on active treatment were rolled over to a rollover study to continue their treatment.
Groups:
- Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine): Participants with non-squamous NSCLC will receive chemotherapy with pemetrexed in combination with either cisplatin or carboplatin (per investigator discretion) on Day 1 of each 21-day cycle for 4 or 6 cycles as per local standard of care, followed by maintenance therapy with pemetrexed alone as per local standard of care until disease progression (per RECIST v1.1), unacceptable toxicity, or death (maximum up to approximately 58 months).
  Participants with squamous NSCLC will receive chemotherapy with gemcitabine on Days 1 and 8 of each 21-day cycle in combination with either cisplatin or carboplatin on Day 1 of each 21-day cycle for 4 or 6 cycles as per local standard of care, followed by best supportive care as per local standard of care until disease progression, unacceptable toxicity, or death (maximum up to approximately 58 months).
Period: Overall Study
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Started | 287 | 285
Completed | 0 | 0
Not Completed | 287 | 285
Not completed — Death | 211 | 201
Not completed — Withdrawal by Subject | 24 | 17
Not completed — Study Terminated By Sponsor | 48 | 59
Not completed — Lost to Follow-up | 3 | 5
Not completed — Local ethics requires subjects' data be removed from aug 2020 to currently. | 0 | 1
Not completed — Participant Moved Into Roll-Over Study | 0 | 2
Not completed — Sponsor Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab | Total
Number analyzed (Participants) | 287 | 285 | 572
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.8 (8.8) | 63.1 (8.8) | 63.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 87 | 176
  Male | 198 | 198 | 396
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 21 | 35
  Not Hispanic or Latino | 265 | 262 | 527
  Unknown or Not Reported | 8 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 33 | 48 | 81
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 247 | 232 | 479
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in the TC3 or IC3-WT Populations
Description: OS is defined as the time from randomization to death from any cause.
Time Frame: From randomization to death from any cause until data cut-off on 10 September 2018 (up to approximately 38 months)
Population: Analysis was performed for the TC3 or IC3-WT populations. Comparison of the treatment arms was performed in randomized participants who were selected on the basis of a minimum level of PD-L1 expression on tumor cells (TCs) and/or immune cells (ICs) with populations excluding participants with a sensitizing EGFR mutation or ALK translocation (i.e., wild type [WT]).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 98 | 107
Months | 13.1 [7.4 to 16.5] | 20.2 [16.5 to NA] — Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events.
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; TC3 or IC3-WT Population; Test type: Superiority — Stratified analysis. OS was tested hierarchically in the efficacy analysis populations; p = 0.0106, Log Rank; Hazard Ratio (HR) = 0.595, 95% CI 2-sided [0.398 to 0.890]

2. Primary Outcome: Overall Survival (OS) in the TC2/3 or IC2/3-WT and TC1/2/3 or IC1/2/3-WT Populations
Description: OS is defined as the time from randomization to death from any cause.
Time Frame: From randomization to death from any cause until data cut-off on 4 February 2020 (up to approximately 54.5 months)
Population: Analysis was performed for the TC2/3 or IC2/3-WT and TC1/2/3 or IC1/2/3-WT populations. Comparison of the treatment arms was performed in randomized participants who were selected on the basis of a minimum level of PD-L1 expression on tumor cells (TCs) and/or immune cells (ICs) with populations excluding participants with a sensitizing EGFR mutation or ALK translocation (i.e., wild type [WT]).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 277 | 277
Months
  TC2/3 or IC2/3-WT Population: number analyzed (Participants) | 162 | 166
  TC2/3 or IC2/3-WT Population | 16.1 [12.6 to 18.0] | 19.9 [17.2 to 25.3]
  TC1/2/3 or IC1/2/3-WT Population | 14.7 [11.2 to 16.5] | 18.9 [13.4 to 23.0]
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; TC2/3 or IC2/3-WT Population; Test type: Superiority — Stratified analysis. OS was tested hierarchically in the efficacy analysis populations; p = 0.3091, Log Rank; Hazard Ratio (HR) = 0.868, 95% CI 2-sided [0.661 to 1.140]
Statistical Analysis 2: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; TC1/2/3 or IC/1/2/3-WT; Test type: Superiority — Stratified analysis. OS was tested hierarchically in the efficacy analysis populations; p = 0.1070, Log Rank — P-value is descriptive as it was not formally tested; Hazard Ratio (HR) = 0.845, 95% CI 2-sided [0.688 to 1.037]

3. Secondary Outcome: Progression-free Survival (PFS) in the TC3 or IC3-WT Populations
Description: PFS is defined as the time from randomization to the first occurrence of disease progression, as determined by the investigator with use of RECIST v1.1, or death from any cause, whichever occurs first. PFS could not be formally tested.
Time Frame: From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first until data cut-off on 10 September 2018 (up to approximately 38 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 98 | 107
Months | 5.0 [4.2 to 5.7] | 8.1 [6.8 to 11.0]
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; TC3 or IC3-WT Population; Test type: Superiority — Stratified Analysis; p = 0.0070, Log Rank — P-value is descriptive as it was not formally tested; Hazard Ratio (HR) = 0.630, 95% CI 2-sided [0.449 to 0.884]

4. Secondary Outcome: Progression-free Survival (PFS) in the TC2/3 or IC2/3-WT and TC1/2/3 or IC1/2/3-WT Populations
Description: as for outcome 3
Time Frame: From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first until data cut-off on 4 February 2020 (up to approximately 54.5 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 277 | 277
Months
  TC2/3 or IC2/3-WT Population: number analyzed (Participants) | 162 | 166
  TC2/3 or IC2/3-WT Population | 5.5 [4.5 to 5.7] | 7.3 [5.6 to 9.3]
  TC1/2/3 or IC1/2/3-WT Population | 5.6 [4.7 to 5.7] | 5.8 [5.5 to 7.3]
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine); TC2/3 or IC2/3-WT Population; Test type: Superiority — Stratified Analysis; p = 0.0004, Log Rank — P-value is descriptive as it was not formally tested; Hazard Ratio (HR) = 0.641, 95% CI 2-sided [0.501 to 0.820]
Statistical Analysis 2: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; TC1/2/3 or IC1/2/3-WT Population; Test type: Superiority — Stratified Analysis; p = 0.0004, Log Rank — P-value is descriptive as it was not formally tested; Hazard Ratio (HR) = 0.716, 95% CI 2-sided [0.595 to 0.863]

5. Secondary Outcome: Percentage of Participants With Objective Response (ORR) in the TC3 or IC3-WT Populations
Description: Objective response (partial response plus complete response) as determined by the investigator according to RECIST v1.1.
Time Frame: Every 6 weeks for 48 weeks following Day 1, thereafter every 9 weeks after completion of Week 48 tumor assessment, regardless of treatment delays, until radiographic disease progression until data cut-off on 10 Sep 2018 (up to approximately 38 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 98 | 107
Percentage of participants | 28.6 | 38.3
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; TC3 or IC3-WT Population; Test type: Superiority — Stratified Analysis; Difference in ORR = 9.75, 95% CI 2-sided [-4.07 to 23.56]

6. Secondary Outcome: Percentage of Participants With Objective Response (ORR) in the TC2/3 or IC2/3-WT and TC1/2/3 or IC1/2/3-WT Populations
Description: Objective response (partial response plus complete response) as determined by the investigator according to RECIST v1.1.
Time Frame: Every 6 weeks for 48 weeks following Day 1, thereafter every 9 weeks after completion of Week 48 tumor assessment, regardless of treatment delays, until radiographic disease progression until data cut-off on 4 Feb 2020 (up to approximately 54.5 months)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 277 | 277
Percentage of participants
  TC2/3 or IC2/3-WT Population: number analyzed (Participants) | 162 | 166
  TC2/3 or IC2/3-WT Population | 32.1 | 33.7
  TC1/2/3 or IC1/2/3-WT Population | 32.1 | 31.4
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; TC2/3 or IC2/3-WT Population; Test type: Superiority — Stratified analysis; Difference in ORR = 1.64, 95% CI 2-sided [-9.14 to 12.42]
Statistical Analysis 2: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; TC1/2/3 or IC1/2/3-WT Population; Test type: Superiority — Stratified analysis; Difference in ORR = -0.72, 95% CI 2-sided [-8.84 to 7.39]

7. Secondary Outcome: Duration of Response (DOR) in the TC3 or IC3-WT Populations
Description: DOR is defined as the time from the first occurrence of a documented objective response to the time of disease progression, as determined by the investigator with use of RECIST v1.1, or death from any cause, whichever occurs first.
Time Frame: From first occurrence of a complete response or partial response, whichever occurs first, until first date that progressive disease or death is documented, whichever occurs first until data cut-off on 10 September 2018 (up to approximately 38 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 28 | 41
Months | 6.7 [5.5 to 17.3] | NA [11.8 to NA] — Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events.
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; TC3 or IC3-WT Population; Test type: Superiority — Stratified Analysis; Hazard Ratio (HR) = 0.365, 95% CI 2-sided [0.166 to 0.800]

8. Secondary Outcome: Duration of Response (DOR) in the TC2/3 or IC2/3-WT and TC1/2/3 or IC1/2/3-WT Populations
Description: as for outcome 7
Time Frame: From first occurrence of a complete response or partial response, whichever occurs first, until first date that progressive disease or death is documented, whichever occurs first until data cut-off on 4 February 2020 (up to approximately 54.5 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 89 | 87
Months
  TC2/3 or IC2/3-WT Population: number analyzed (Participants) | 52 | 56
  TC2/3 or IC2/3-WT Population | 5.8 [5.1 to 9.8] | 38.9 [16.9 to NA] — Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events.
  TC1/2/3 or IC1/2/3-WT Population | 5.7 [5.1 to 8.8] | 26.3 [16.1 to 43.7]
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; TC2/3 or IC2/3-WT Population; Test type: Superiority — Stratified analysis; Hazard Ratio (HR) = 0.235, 95% CI 2-sided [0.135 to 0.409]
Statistical Analysis 2: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; TC1/2/3 or IC1/2/3-WT Population; Test type: Superiority — Stratified analysis; Hazard Ratio (HR) = 0.284, 95% CI 2-sided [0.190 to 0.424]

9. Secondary Outcome: Percentage of Participants Who Are Alive at 1 Year in the TC3 or IC3-WT Populations
Time Frame: Baseline to 1 year or death, whichever occurs first until data cut-off on 10 September 2018 (up to approximately 38 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 98 | 107
Percentage of participants | 50.64 [40.00 to 61.27] | 64.90 [55.36 to 74.43]
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; 1-Year TC3 or IC3-WT Population; Test type: Superiority; Difference in Event Free Rate = 14.26, 95% CI 2-sided [-0.03 to 28.55]

10. Secondary Outcome: Percentage of Participants Who Are Alive at 2 Years in the TC3 or IC3-WT Populations
Time Frame: Baseline to 2 years or death, whichever occurs first until data cut-off on 10 September 2018 (up to approximately 38 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 98 | 107
Percentage of participants | 24.79 [13.11 to 36.47] | 45.49 [32.11 to 58.88]
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; 2-Years TC3 or IC3-WT Population; Test type: Superiority; Difference in Event Free Rate = 20.70, 95% CI 2-sided [2.94 to 38.47]

11. Secondary Outcome: Percentage of Participants Who Are Alive at 1 Year in the TC2/3 or IC2/3-WT and TC1/2/3 or IC1/2/3-WT Populations
Time Frame: Baseline to 1 year or death, whichever occurs first until clinical cut-off date on 4 February 2020 (up to approximately 54.5 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 277 | 277
Percentage of participants
  1-Year TC2/3 or IC2/3-WT Population: number analyzed (Participants) | 162 | 166
  1-Year TC2/3 or IC2/3-WT Population | 58.65 [50.95 to 66.35] | 63.39 [56.00 to 70.77]
  1-Year TC1/2/3 or IC1/2/3-WT Population | 54.89 [48.93 to 60.84] | 59.95 [54.12 to 65.78]
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; 1-Year TC2/3 or IC2/3-WT Population; Test type: Superiority; Difference in Event Free Rate = 4.74, 95% CI 2-sided [-5.93 to 15.40]
Statistical Analysis 2: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; 1-Year TC1/2/3 or IC1/2/3-WT Population; Test type: Superiority; Difference in Event Free Rate = 5.06, 95% CI 2-sided [-3.27 to 13.40]

12. Secondary Outcome: Percentage of Participants Who Are Alive at 2 Years in the TC2/3 or IC2/3-WT and TC1/2/3 or IC1/2/3-WT Populations
Time Frame: Baseline to 2 years or death, whichever occurs first until clinical cut-off date on 4 February 2020 (up to approximately 54.5 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 277 | 277
Percentage of participants
  2-Years TC2/3 or IC2/3-WT Population: number analyzed (Participants) | 162 | 166
  2-Years TC2/3 or IC2/3-WT Population | 35.42 [27.91 to 42.94] | 44.15 [36.51 to 51.80]
  2-Years TC1/2/3 or IC1/2/3-WT Population | 30.82 [25.28 to 36.36] | 41.76 [35.84 to 47.67]
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; 2-Years TC2/3 or IC2/3-WT Population; Test type: Superiority; Difference in Event Free Rate = 8.73, 95% CI 2-sided [-1.99 to 19.45]
Statistical Analysis 2: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; 2-Years TC1/2/3 or IC1/2/3-WT Population; Test type: Superiority; Difference in Event Free Rate = 10.94, 95% CI 2-sided [2.83 to 19.04]

13. Secondary Outcome: Time to Deterioration (TTD) in Patient-reported Lung Cancer Symptoms Score as Assessed by the Symptoms in Lung Cancer (SILC) Scale Symptom Score in the TC3 or IC3-WT Populations
Description: TTD in each of the patient-reported lung cancer symptoms with use of the SILC scale. The SILC scale is a nine-item content valid self-report measure of lung cancer symptoms. It measures severity of cough, dyspnea, and chest pain with a total symptom severity score. Each SILC symptom scale (dyspnea, cough, chest pain) score was calculated as the average of the component items (range 0 to 4). An increase in score suggested worsening in symptomatology. A symptom score change of 0.3 points for the dyspnea and cough scores was considered to be clinically significant; whereas a symptom score change of 0.5 points for the chest pain score was considered to be clinically significant.
Time Frame: Baseline until data cut-off on 10 September 2018 (up to approximately 38 months)
Population: Analysis was performed for the TC3 or IC3-WT Populations.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 98 | 107
Months
  Cough | 3.4 [1.3 to 12.4] | 3.5 [1.0 to 10.8]
  Dyspnea | 1.0 [0.5 to 1.9] | 1.3 [0.7 to 3.6]
  Chest pain | 1.1 [0.7 to NA] — Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events. | 1.7 [0.7 to 4.5]
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; Cough in TC3 or IC3-WT Populations; Test type: Superiority — Stratified Analysis; Hazard Ratio (HR) = 1.142, 95% CI 2-sided [0.657 to 1.984]
Statistical Analysis 2: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; Dyspnoea in TC3 or IC3-WT Populations; Test type: Superiority — Stratified analysis; Hazard Ratio (HR) = 0.891, 95% CI 2-sided [0.555 to 1.430]
Statistical Analysis 3: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; Chest pain in TC3 or IC3-WT Populations; Test type: Superiority — Stratified analysis; Hazard Ratio (HR) = 1.229, 95% CI 2-sided [0.737 to 2.049]

14. Secondary Outcome: Change From Baseline in Patient-reported Lung Cancer Symptoms Score as Assessed by the SILC Scale Symptom Score in the TC3 or IC3-WT Populations
Description: Change from baseline in each of the patient-reported lung cancer symptoms with use of the SILC scale. The SILC scale is a nine-item content valid self-report measure of lung cancer symptoms. It measures severity of cough, dyspnea, and chest pain with a total symptom severity score. Each SILC symptom scale (dyspnea, cough, chest pain) score was calculated as the average of the component items (range 0 to 4). An increase in score suggested worsening in symptomatology. A symptom score change of 0.3 points for the dyspnea and cough scores was considered to be clinically significant; whereas a symptom score change of 0.5 points for the chest pain score was considered to be clinically significant.
Time Frame: Baseline until data cut-off on 10 September 2018 (up to approximately 38 months)
Population: Analysis was performed for the TC3 or IC3-WT Populations.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 52 | 61
Score on a scale
  Chest Pain, Week 1: number analyzed (Participants) | 44 | 47
  Chest Pain, Week 1 | 0.57 (1.23) | 0.31 (0.84)
  Chest Pain, Week 2: number analyzed (Participants) | 42 | 48
  Chest Pain, Week 2 | 0.42 (1.13) | 0.33 (0.85)
  Chest Pain, Week 3: number analyzed (Participants) | 44 | 49
  Chest Pain, Week 3 | 0.25 (1.26) | 0.43 (0.97)
  Chest Pain, Week 4: number analyzed (Participants) | 41 | 49
  Chest Pain, Week 4 | 0.15 (1.21) | 0.43 (1.08)
  Chest Pain, Week 5: number analyzed (Participants) | 39 | 47
  Chest Pain, Week 5 | 0.27 (1.19) | 0.28 (1.00)
  Chest Pain, Week 6: number analyzed (Participants) | 33 | 48
  Chest Pain, Week 6 | 0.30 (1.26) | 0.25 (0.85)
  Chest Pain, Week 7: number analyzed (Participants) | 30 | 44
  Chest Pain, Week 7 | 0.23 (1.04) | 0.30 (0.97)
  Chest Pain, Week 8: number analyzed (Participants) | 29 | 44
  Chest Pain, Week 8 | 0.17 (1.12) | 0.20 (0.82)
  Chest Pain, Week 9: number analyzed (Participants) | 31 | 47
  Chest Pain, Week 9 | 0.27 (1.00) | 0.33 (1.07)
  Chest Pain, Week 10: number analyzed (Participants) | 30 | 40
  Chest Pain, Week 10 | 0.30 (1.13) | 0.25 (1.12)
  Chest Pain, Week 11: number analyzed (Participants) | 29 | 34
  Chest Pain, Week 11 | 0.26 (1.32) | 0.21 (0.96)
  Chest Pain, Week 12: number analyzed (Participants) | 32 | 40
  Chest Pain, Week 12 | 0.22 (1.33) | 0.33 (0.97)
  Chest Pain, Week 13: number analyzed (Participants) | 28 | 38
  Chest Pain, Week 13 | 0.07 (1.17) | 0.30 (1.04)
  Chest Pain, Week 14: number analyzed (Participants) | 28 | 35
  Chest Pain, Week 14 | 0.07 (1.16) | 0.27 (0.85)
  Chest Pain, Week 15: number analyzed (Participants) | 30 | 40
  Chest Pain, Week 15 | 0.10 (1.23) | 0.45 (1.01)
  Chest Pain, Week 16: number analyzed (Participants) | 25 | 32
  Chest Pain, Week 16 | 0.00 (1.20) | 0.19 (0.99)
  Chest Pain, Week 17: number analyzed (Participants) | 27 | 34
  Chest Pain, Week 17 | 0.22 (1.41) | 0.22 (1.20)
  Chest Pain, Week 18: number analyzed (Participants) | 23 | 37
  Chest Pain, Week 18 | 0.11 (1.26) | 0.26 (0.85)
  Chest Pain, Week 19: number analyzed (Participants) | 22 | 32
  Chest Pain, Week 19 | 0.11 (1.01) | 0.23 (0.94)
  Chest Pain, Week 20: number analyzed (Participants) | 22 | 35
  Chest Pain, Week 20 | 0.20 (1.32) | 0.23 (0.95)
  Chest Pain, Week 21: number analyzed (Participants) | 18 | 36
  Chest Pain, Week 21 | 0.03 (0.83) | 0.11 (0.87)
  Chest Pain, Week 22: number analyzed (Participants) | 20 | 35
  Chest Pain, Week 22 | 0.30 (1.35) | 0.19 (1.02)
  Chest Pain, Week 23: number analyzed (Participants) | 16 | 33
  Chest Pain, Week 23 | 0.00 (1.00) | 0.33 (0.84)
  Chest Pain, Week 24: number analyzed (Participants) | 16 | 33
  Chest Pain, Week 24 | -0.09 (0.88) | 0.18 (1.13)
  Chest Pain, Week 25: number analyzed (Participants) | 11 | 29
  Chest Pain, Week 25 | 0.27 (0.79) | 0.29 (0.87)
  Chest Pain, Week 26: number analyzed (Participants) | 13 | 32
  Chest Pain, Week 26 | 0.12 (1.31) | 0.11 (0.72)
  Chest Pain, Week 27: number analyzed (Participants) | 11 | 32
  Chest Pain, Week 27 | 0.05 (1.15) | 0.20 (0.80)
  Chest Pain, Week 28: number analyzed (Participants) | 11 | 30
  Chest Pain, Week 28 | 0.00 (0.81) | 0.23 (0.98)
  Chest Pain, Week 29: number analyzed (Participants) | 12 | 28
  Chest Pain, Week 29 | -0.25 (0.87) | 0.18 (0.80)
  Chest Pain, Week 30: number analyzed (Participants) | 12 | 30
  Chest Pain, Week 30 | 0.21 (1.45) | 0.32 (0.95)
  Chest Pain, Week 31: number analyzed (Participants) | 11 | 29
  Chest Pain, Week 31 | 0.18 (1.72) | 0.33 (0.90)
  Chest Pain, Week 32: number analyzed (Participants) | 11 | 23
  Chest Pain, Week 32 | 0.41 (1.61) | 0.35 (1.20)
  Chest Pain, Week 33: number analyzed (Participants) | 13 | 26
  Chest Pain, Week 33 | 0.00 (1.44) | 0.04 (1.03)
  Chest Pain, Week 34: number analyzed (Participants) | 10 | 26
  Chest Pain, Week 34 | 0.40 (1.31) | 0.31 (0.98)
  Chest Pain, Week 35: number analyzed (Participants) | 11 | 27
  Chest Pain, Week 35 | 0.00 (1.16) | 0.28 (1.13)
  Chest Pain, Week 36: number analyzed (Participants) | 9 | 25
  Chest Pain, Week 36 | 0.06 (0.85) | 0.08 (0.95)
  Chest Pain, Week 37: number analyzed (Participants) | 8 | 23
  Chest Pain, Week 37 | 0.31 (1.25) | 0.39 (0.89)
  Chest Pain, Week 38: number analyzed (Participants) | 11 | 21
  Chest Pain, Week 38 | 0.23 (0.72) | 0.31 (1.20)
  Chest Pain, Week 39: number analyzed (Participants) | 9 | 22
  Chest Pain, Week 39 | 0.22 (1.00) | 0.14 (0.92)
  Chest Pain, Week 40: number analyzed (Participants) | 7 | 23
  Chest Pain, Week 40 | 0.43 (1.02) | 0.30 (1.21)
  Chest Pain, Week 41: number analyzed (Participants) | 7 | 20
  Chest Pain, Week 41 | 0.36 (1.07) | 0.30 (1.01)
  Chest Pain, Week 42: number analyzed (Participants) | 6 | 20
  Chest Pain, Week 42 | 0.25 (1.04) | 0.33 (1.05)
  Chest Pain, Week 43: number analyzed (Participants) | 5 | 20
  Chest Pain, Week 43 | 0.30 (1.15) | 0.18 (1.29)
  Chest Pain, Week 44: number analyzed (Participants) | 7 | 19
  Chest Pain, Week 44 | 0.14 (0.99) | 0.42 (1.15)
  Chest Pain, Week 45: number analyzed (Participants) | 4 | 21
  Chest Pain, Week 45 | 0.63 (0.48) | 0.31 (0.90)
  Chest Pain, Week 46: number analyzed (Participants) | 5 | 19
  Chest Pain, Week 46 | 0.30 (0.45) | 0.37 (0.93)
  Chest Pain, Week 47: number analyzed (Participants) | 4 | 18
  Chest Pain, Week 47 | 0.50 (0.71) | 0.31 (0.86)
  Chest Pain, Week 48: number analyzed (Participants) | 3 | 15
  Chest Pain, Week 48 | 0.50 (0.50) | 0.17 (0.79)
  Chest Pain, Week 49: number analyzed (Participants) | 3 | 17
  Chest Pain, Week 49 | 1.00 (1.32) | 0.47 (1.07)
  Chest Pain, Week 50: number analyzed (Participants) | 5 | 15
  Chest Pain, Week 50 | 0.80 (0.91) | 0.20 (0.92)
  Chest Pain, Week 51: number analyzed (Participants) | 4 | 16
  Chest Pain, Week 51 | 0.88 (0.85) | 0.31 (0.89)
  Chest Pain, Week 52: number analyzed (Participants) | 4 | 13
  Chest Pain, Week 52 | 0.75 (1.19) | 0.54 (1.11)
  Chest Pain, Week 53: number analyzed (Participants) | 5 | 12
  Chest Pain, Week 53 | 0.70 (0.84) | 0.29 (1.08)
  Chest Pain, Week 54: number analyzed (Participants) | 4 | 14
  Chest Pain, Week 54 | 1.13 (1.03) | 0.25 (0.87)
  Chest Pain, Week 55: number analyzed (Participants) | 3 | 13
  Chest Pain, Week 55 | 1.17 (1.26) | 0.15 (0.99)
  Chest Pain, Week 56: number analyzed (Participants) | 4 | 14
  Chest Pain, Week 56 | 0.38 (0.48) | 0.29 (0.96)
  Chest Pain, Week 57: number analyzed (Participants) | 3 | 13
  Chest Pain, Week 57 | 0.67 (0.58) | 0.08 (0.73)
  Chest Pain, Week 58: number analyzed (Participants) | 3 | 13
  Chest Pain, Week 58 | 1.17 (1.04) | 0.19 (1.07)
  Chest Pain, Week 59: number analyzed (Participants) | 3 | 9
  Chest Pain, Week 59 | 1.00 (0.87) | 0.00 (0.87)
  Chest Pain, Week 60: number analyzed (Participants) | 2 | 13
  Chest Pain, Week 60 | 0.50 (1.41) | 0.38 (1.08)
  Chest Pain, Week 61: number analyzed (Participants) | 3 | 14
  Chest Pain, Week 61 | 1.00 (0.87) | 0.36 (1.12)
  Chest Pain, Week 62: number analyzed (Participants) | 3 | 14
  Chest Pain, Week 62 | 0.83 (0.76) | 0.43 (1.16)
  Chest Pain, Week 63: number analyzed (Participants) | 2 | 12
  Chest Pain, Week 63 | 0.50 (0.71) | 0.29 (0.86)
  Chest Pain, Week 64: number analyzed (Participants) | 1 | 10
  Chest Pain, Week 64 | 0.00 | 0.40 (1.22)
  Chest Pain, Week 65: number analyzed (Participants) | 1 | 13
  Chest Pain, Week 65 | 0.00 | 0.35 (1.11)
  Chest Pain, Week 66: number analyzed (Participants) | 1 | 11
  Chest Pain, Week 66 | 0.00 | 0.45 (1.44)
  Chest Pain, Week 67: number analyzed (Participants) | 2 | 11
  Chest Pain, Week 67 | 1.00 (1.41) | -0.09 (0.80)
  Chest Pain, Week 68: number analyzed (Participants) | 2 | 9
  Chest Pain, Week 68 | 0.75 (1.06) | 0.39 (1.45)
  Chest Pain, Week 69: number analyzed (Participants) | 2 | 10
  Chest Pain, Week 69 | 0.50 (0.71) | 0.50 (1.33)
  Chest Pain, Week 70: number analyzed (Participants) | 2 | 11
  Chest Pain, Week 70 | 1.00 (1.41) | 0.18 (0.81)
  Chest Pain, Week 71: number analyzed (Participants) | 2 | 10
  Chest Pain, Week 71 | 0.50 (0.71) | 0.45 (1.32)
  Chest Pain, Week 72: number analyzed (Participants) | 1 | 12
  Chest Pain, Week 72 | 1.00 | 0.42 (1.18)
  Chest Pain, Week 73: number analyzed (Participants) | 1 | 11
  Chest Pain, Week 73 | 1.50 | 0.27 (1.19)
  Chest Pain, Week 74: number analyzed (Participants) | 2 | 9
  Chest Pain, Week 74 | 0.50 (0.71) | 0.50 (1.30)
  Chest Pain, Week 75: number analyzed (Participants) | 2 | 9
  Chest Pain, Week 75 | 0.75 (1.06) | 0.33 (1.32)
  Chest Pain, Week 76: number analyzed (Participants) | 2 | 8
  Chest Pain, Week 76 | 0.50 (0.71) | 0.00 (0.93)
  Chest Pain, Week 77: number analyzed (Participants) | 2 | 8
  Chest Pain, Week 77 | 0.50 (0.71) | 0.19 (1.33)
  Chest Pain, Week 78: number analyzed (Participants) | 2 | 7
  Chest Pain, Week 78 | 1.00 (1.41) | 0.21 (1.44)
  Chest Pain, Week 79: number analyzed (Participants) | 2 | 8
  Chest Pain, Week 79 | 0.50 (0.71) | 0.31 (1.31)
  Chest Pain, Week 80: number analyzed (Participants) | 2 | 9
  Chest Pain, Week 80 | 0.75 (1.06) | 0.72 (1.70)
  Chest Pain, Week 81: number analyzed (Participants) | 2 | 6
  Chest Pain, Week 81 | 0.75 (1.06) | 0.08 (1.72)
  Chest Pain, Week 82: number analyzed (Participants) | 1 | 6
  Chest Pain, Week 82 | 0.00 | 0.08 (1.24)
  Chest Pain, Week 83: number analyzed (Participants) | 1 | 6
  Chest Pain, Week 83 | 0.00 | 0.50 (1.48)
  Chest Pain, Week 84: number analyzed (Participants) | 1 | 7
  Chest Pain, Week 84 | 0.50 | 0.43 (1.43)
  Chest Pain, Week 85: number analyzed (Participants) | 1 | 8
  Chest Pain, Week 85 | 0.00 | 0.38 (1.41)
  Chest Pain, Week 86: number analyzed (Participants) | 1 | 7
  Chest Pain, Week 86 | 0.00 | 0.21 (1.44)
  Chest Pain, Week 87: number analyzed (Participants) | 1 | 7
  Chest Pain, Week 87 | 0.00 | 0.29 (1.41)
  Chest Pain, Week 88: number analyzed (Participants) | 0 | 7
  Chest Pain, Week 88 |  | 0.43 (1.17)
  Chest Pain, Week 89: number analyzed (Participants) | 0 | 5
  Chest Pain, Week 89 |  | -0.20 (0.91)
  Chest Pain, Week 90: number analyzed (Participants) | 0 | 7
  Chest Pain, Week 90 |  | 0.07 (1.13)
  Chest Pain, Week 91: number analyzed (Participants) | 0 | 7
  Chest Pain, Week 91 |  | -0.07 (0.89)
  Chest Pain, Week 92: number analyzed (Participants) | 0 | 6
  Chest Pain, Week 92 |  | 0.33 (1.54)
  Chest Pain, Week 93: number analyzed (Participants) | 0 | 7
  Chest Pain, Week 93 |  | 0.50 (1.47)
  Chest Pain, Week 94: number analyzed (Participants) | 0 | 5
  Chest Pain, Week 94 |  | 0.20 (1.35)
  Chest Pain, Week 95: number analyzed (Participants) | 0 | 6
  Chest Pain, Week 95 |  | 0.33 (1.54)
  Chest Pain, Week 96: number analyzed (Participants) | 0 | 6
  Chest Pain, Week 96 |  | 0.33 (1.54)
  Chest Pain, Week 97: number analyzed (Participants) | 0 | 7
  Chest Pain, Week 97 |  | 0.50 (1.47)
  Chest Pain, Week 98: number analyzed (Participants) | 0 | 6
  Chest Pain, Week 98 |  | 0.33 (1.54)
  Chest Pain, Week 99: number analyzed (Participants) | 0 | 4
  Chest Pain, Week 99 |  | 0.88 (1.18)
  Chest Pain, Week 100: number analyzed (Participants) | 0 | 5
  Chest Pain, Week 100 |  | 0.50 (1.00)
  Chest Pain, Week 101: number analyzed (Participants) | 0 | 6
  Chest Pain, Week 101 |  | 0.83 (0.93)
  Chest Pain, Week 102: number analyzed (Participants) | 0 | 5
  Chest Pain, Week 102 |  | 0.50 (1.00)
  Chest Pain, Week 103: number analyzed (Participants) | 0 | 4
  Chest Pain, Week 103 |  | 0.63 (1.11)
  Chest Pain, Week 104: number analyzed (Participants) | 0 | 3
  Chest Pain, Week 104 |  | 1.00 (1.00)
  Chest Pain, Week 105: number analyzed (Participants) | 0 | 3
  Chest Pain, Week 105 |  | 1.00 (1.00)
  Chest Pain, Week 106: number analyzed (Participants) | 0 | 2
  Chest Pain, Week 106 |  | 0.50 (0.71)
  Chest Pain, Week 107: number analyzed (Participants) | 0 | 3
  Chest Pain, Week 107 |  | 1.00 (1.00)
  Chest Pain, Week 108: number analyzed (Participants) | 0 | 2
  Chest Pain, Week 108 |  | 1.50 (0.71)
  Chest Pain, Week 109: number analyzed (Participants) | 0 | 2
  Chest Pain, Week 109 |  | 1.75 (1.06)
  Chest Pain, Week 110: number analyzed (Participants) | 0 | 2
  Chest Pain, Week 110 |  | 2.00 (1.41)
  Chest Pain, Week 111: number analyzed (Participants) | 0 | 2
  Chest Pain, Week 111 |  | 1.50 (0.71)
  Chest Pain, Week 112: number analyzed (Participants) | 0 | 2
  Chest Pain, Week 112 |  | 1.50 (0.71)
  Chest Pain, Week 113: number analyzed (Participants) | 0 | 2
  Chest Pain, Week 113 |  | 1.50 (0.71)
  Chest Pain, Week 114: number analyzed (Participants) | 0 | 2
  Chest Pain, Week 114 |  | 2.00 (1.41)
  Chest Pain, Week 115: number analyzed (Participants) | 0 | 2
  Chest Pain, Week 115 |  | 1.75 (1.06)
  Chest Pain, Week 116: number analyzed (Participants) | 0 | 2
  Chest Pain, Week 116 |  | 2.00 (1.41)
  Chest Pain, Week 117: number analyzed (Participants) | 0 | 2
  Chest Pain, Week 117 |  | 2.00 (1.41)
  Chest Pain, Week 118: number analyzed (Participants) | 0 | 2
  Chest Pain, Week 118 |  | 2.00 (1.41)
  Chest Pain, Week 119: number analyzed (Participants) | 0 | 2
  Chest Pain, Week 119 |  | 1.75 (1.06)
  Chest Pain, Week 120: number analyzed (Participants) | 0 | 1
  Chest Pain, Week 120 |  | 2.50
  Chest Pain, Week 121: number analyzed (Participants) | 0 | 1
  Chest Pain, Week 121 |  | 2.00
  Chest Pain, Week 122: number analyzed (Participants) | 0 | 1
  Chest Pain, Week 122 |  | 3.00
  Chest Pain, Week 123: number analyzed (Participants) | 0 | 1
  Chest Pain, Week 123 |  | 2.50
  Chest Pain, Week 124: number analyzed (Participants) | 0 | 1
  Chest Pain, Week 124 |  | 3.00
  Chest Pain, Week 125: number analyzed (Participants) | 0 | 1
  Chest Pain, Week 125 |  | 3.00
  Chest Pain, Week 126: number analyzed (Participants) | 0 | 1
  Chest Pain, Week 126 |  | 3.00
  Chest Pain, Week 127: number analyzed (Participants) | 0 | 1
  Chest Pain, Week 127 |  | 2.00
  Chest Pain, Week 128: number analyzed (Participants) | 0 | 1
  Chest Pain, Week 128 |  | 3.00
  Chest Pain, Week 129: number analyzed (Participants) | 0 | 1
  Chest Pain, Week 129 |  | 3.00
  Chest Pain, Week 130: number analyzed (Participants) | 0 | 1
  Chest Pain, Week 130 |  | 2.00
  Chest Pain, Week 131: number analyzed (Participants) | 0 | 1
  Chest Pain, Week 131 |  | 2.00
  Cough, Week 1: number analyzed (Participants) | 44 | 47
  Cough, Week 1 | 0.13 (0.86) | 0.10 (0.70)
  Cough, Week 2: number analyzed (Participants) | 42 | 48
  Cough, Week 2 | -0.01 (0.99) | 0.19 (0.75)
  Cough, Week 3: number analyzed (Participants) | 44 | 49
  Cough, Week 3 | -0.03 (0.76) | -0.01 (0.76)
  Cough, Week 4: number analyzed (Participants) | 41 | 49
  Cough, Week 4 | -0.02 (1.02) | -0.03 (0.98)
  Cough, Week 5: number analyzed (Participants) | 39 | 47
  Cough, Week 5 | -0.01 (0.84) | 0.00 (0.96)
  Cough, Week 6: number analyzed (Participants) | 33 | 48
  Cough, Week 6 | -0.18 (0.93) | -0.18 (0.89)
  Cough, Week 7: number analyzed (Participants) | 30 | 44
  Cough, Week 7 | -0.20 (0.92) | -0.06 (0.98)
  Cough, Week 8: number analyzed (Participants) | 29 | 44
  Cough, Week 8 | -0.10 (0.90) | -0.13 (0.91)
  Cough, Week 9: number analyzed (Participants) | 31 | 47
  Cough, Week 9 | -0.24 (0.86) | -0.06 (1.01)
  Cough, Week 10: number analyzed (Participants) | 30 | 40
  Cough, Week 10 | -0.07 (1.12) | -0.10 (1.02)
  Cough, Week 11: number analyzed (Participants) | 29 | 34
  Cough, Week 11 | 0.02 (1.24) | -0.07 (1.07)
  Cough, Week 12: number analyzed (Participants) | 32 | 40
  Cough, Week 12 | -0.08 (1.30) | -0.09 (0.97)
  Cough, Week 13: number analyzed (Participants) | 28 | 38
  Cough, Week 13 | -0.09 (1.22) | -0.20 (0.93)
  Cough, Week 14: number analyzed (Participants) | 28 | 35
  Cough, Week 14 | -0.20 (1.19) | -0.07 (0.95)
  Cough, Week 15: number analyzed (Participants) | 30 | 40
  Cough, Week 15 | -0.05 (1.35) | -0.19 (1.04)
  Cough, Week 16: number analyzed (Participants) | 25 | 32
  Cough, Week 16 | -0.10 (1.06) | -0.19 (0.94)
  Cough, Week 17: number analyzed (Participants) | 27 | 34
  Cough, Week 17 | -0.04 (0.99) | -0.21 (1.09)
  Cough, Week 18: number analyzed (Participants) | 23 | 37
  Cough, Week 18 | 0.02 (1.23) | -0.26 (0.93)
  Cough, Week 19: number analyzed (Participants) | 22 | 32
  Cough, Week 19 | -0.23 (1.29) | -0.27 (0.87)
  Cough, Week 20: number analyzed (Participants) | 22 | 35
  Cough, Week 20 | 0.00 (1.33) | -0.33 (0.95)
  Cough, Week 21: number analyzed (Participants) | 18 | 36
  Cough, Week 21 | -0.17 (1.40) | -0.19 (0.88)
  Cough, Week 22: number analyzed (Participants) | 20 | 35
  Cough, Week 22 | -0.20 (1.32) | -0.17 (0.89)
  Cough, Week 23: number analyzed (Participants) | 16 | 33
  Cough, Week 23 | -0.22 (1.18) | 0.05 (0.90)
  Cough, Week 24: number analyzed (Participants) | 16 | 33
  Cough, Week 24 | -0.13 (1.51) | -0.12 (0.80)
  Cough, Week 25: number analyzed (Participants) | 11 | 29
  Cough, Week 25 | -0.45 (0.96) | 0.14 (0.82)
  Cough, Week 26: number analyzed (Participants) | 13 | 32
  Cough, Week 26 | -0.46 (1.20) | -0.03 (0.89)
  Cough, Week 27: number analyzed (Participants) | 11 | 32
  Cough, Week 27 | -0.50 (1.22) | -0.05 (0.94)
  Cough, Week 28: number analyzed (Participants) | 11 | 30
  Cough, Week 28 | -0.45 (0.88) | 0.08 (0.84)
  Cough, Week 29: number analyzed (Participants) | 12 | 28
  Cough, Week 29 | -0.50 (1.31) | 0.05 (0.67)
  Cough, Week 30: number analyzed (Participants) | 12 | 30
  Cough, Week 30 | -0.88 (1.13) | 0.12 (0.88)
  Cough, Week 31: number analyzed (Participants) | 11 | 29
  Cough, Week 31 | -0.86 (1.40) | 0.05 (0.74)
  Cough, Week 32: number analyzed (Participants) | 11 | 23
  Cough, Week 32 | -0.73 (1.56) | -0.04 (1.04)
  Cough, Week 33: number analyzed (Participants) | 13 | 26
  Cough, Week 33 | -0.77 (1.13) | -0.29 (1.06)
  Cough, Week 34: number analyzed (Participants) | 10 | 26
  Cough, Week 34 | -0.80 (1.18) | -0.02 (0.75)
  Cough, Week 35: number analyzed (Participants) | 11 | 27
  Cough, Week 35 | -0.14 (0.95) | -0.09 (1.10)
  Cough, Week 36: number analyzed (Participants) | 9 | 25
  Cough, Week 36 | -0.17 (0.66) | -0.36 (1.16)
  Cough, Week 37: number analyzed (Participants) | 8 | 23
  Cough, Week 37 | -0.25 (0.89) | -0.04 (0.84)
  Cough, Week 38: number analyzed (Participants) | 11 | 21
  Cough, Week 38 | 0.05 (0.88) | -0.07 (1.11)
  Cough, Week 39: number analyzed (Participants) | 9 | 22
  Cough, Week 39 | -0.50 (0.90) | -0.20 (0.97)
  Cough, Week 40: number analyzed (Participants) | 7 | 23
  Cough, Week 40 | -0.36 (0.94) | -0.39 (1.23)
  Cough, Week 41: number analyzed (Participants) | 7 | 20
  Cough, Week 41 | 0.21 (0.57) | 0.05 (0.84)
  Cough, Week 42: number analyzed (Participants) | 6 | 20
  Cough, Week 42 | 0.17 (0.52) | -0.20 (1.16)
  Cough, Week 43: number analyzed (Participants) | 5 | 20
  Cough, Week 43 | 0.10 (0.55) | 0.03 (1.06)
  Cough, Week 44: number analyzed (Participants) | 7 | 19
  Cough, Week 44 | 0.36 (0.94) | -0.11 (1.09)
  Cough, Week 45: number analyzed (Participants) | 4 | 21
  Cough, Week 45 | 0.25 (0.50) | -0.26 (0.92)
  Cough, Week 46: number analyzed (Participants) | 5 | 19
  Cough, Week 46 | 0.10 (0.96) | 0.08 (0.85)
  Cough, Week 47: number analyzed (Participants) | 4 | 18
  Cough, Week 47 | 0.50 (0.58) | -0.03 (0.90)
  Cough, Week 48: number analyzed (Participants) | 3 | 15
  Cough, Week 48 | 0.17 (0.29) | 0.23 (0.68)
  Cough, Week 49: number analyzed (Participants) | 3 | 17
  Cough, Week 49 | 0.67 (0.76) | 0.26 (0.85)
  Cough, Week 50: number analyzed (Participants) | 5 | 15
  Cough, Week 50 | 0.30 (0.76) | 0.00 (0.85)
  Cough, Week 51: number analyzed (Participants) | 4 | 16
  Cough, Week 51 | 0.13 (0.63) | 0.06 (0.93)
  Cough, Week 52: number analyzed (Participants) | 4 | 13
  Cough, Week 52 | 0.63 (0.95) | 0.27 (0.97)
  Cough, Week 53: number analyzed (Participants) | 5 | 12
  Cough, Week 53 | 0.70 (0.76) | 0.38 (0.71)
  Cough, Week 54: number analyzed (Participants) | 4 | 14
  Cough, Week 54 | 0.50 (0.41) | 0.07 (0.70)
  Cough, Week 55: number analyzed (Participants) | 3 | 13
  Cough, Week 55 | 0.67 (0.29) | 0.12 (0.94)
  Cough, Week 56: number analyzed (Participants) | 4 | 14
  Cough, Week 56 | 0.50 (0.41) | 0.14 (0.97)
  Cough, Week 57: number analyzed (Participants) | 3 | 13
  Cough, Week 57 | 0.50 (0.50) | 0.15 (0.66)
  Cough, Week 58: number analyzed (Participants) | 3 | 13
  Cough, Week 58 | 0.67 (0.29) | 0.08 (1.00)
  Cough, Week 59: number analyzed (Participants) | 3 | 9
  Cough, Week 59 | 0.33 (0.58) | 0.06 (0.63)
  Cough, Week 60: number analyzed (Participants) | 2 | 13
  Cough, Week 60 | 0.75 (0.35) | -0.04 (0.83)
  Cough, Week 61: number analyzed (Participants) | 3 | 14
  Cough, Week 61 | 0.50 (0.50) | 0.00 (0.88)
  Cough, Week 62: number analyzed (Participants) | 3 | 14
  Cough, Week 62 | 0.33 (0.58) | 0.14 (0.79)
  Cough, Week 63: number analyzed (Participants) | 2 | 12
  Cough, Week 63 | 0.00 (0.00) | -0.04 (0.86)
  Cough, Week 64: number analyzed (Participants) | 1 | 10
  Cough, Week 64 | 0.00 | 0.35 (1.00)
  Cough, Week 65: number analyzed (Participants) | 1 | 13
  Cough, Week 65 | 0.50 | 0.12 (0.92)
  Cough, Week 66: number analyzed (Participants) | 1 | 11
  Cough, Week 66 | 0.00 | 0.45 (1.21)
  Cough, Week 67: number analyzed (Participants) | 2 | 11
  Cough, Week 67 | 0.25 (0.35) | -0.09 (0.66)
  Cough, Week 68: number analyzed (Participants) | 2 | 9
  Cough, Week 68 | 0.25 (0.35) | 0.61 (1.29)
  Cough, Week 69: number analyzed (Participants) | 2 | 10
  Cough, Week 69 | 0.25 (0.35) | 0.50 (1.18)
  Cough, Week 70: number analyzed (Participants) | 2 | 11
  Cough, Week 70 | 0.25 (0.35) | 0.23 (0.79)
  Cough, Week 71: number analyzed (Participants) | 2 | 10
  Cough, Week 71 | 0.00 (0.00) | 0.55 (0.90)
  Cough, Week 72: number analyzed (Participants) | 1 | 12
  Cough, Week 72 | -0.50 | 0.42 (0.93)
  Cough, Week 73: number analyzed (Participants) | 1 | 11
  Cough, Week 73 | 0.00 | 0.64 (1.07)
  Cough, Week 74: number analyzed (Participants) | 2 | 9
  Cough, Week 74 | 0.00 (0.00) | 0.56 (1.04)
  Cough, Week 75: number analyzed (Participants) | 2 | 9
  Cough, Week 75 | 0.00 (0.71) | 0.67 (1.35)
  Cough, Week 76: number analyzed (Participants) | 2 | 8
  Cough, Week 76 | 0.25 (0.35) | 0.31 (1.00)
  Cough, Week 77: number analyzed (Participants) | 2 | 8
  Cough, Week 77 | 0.00 (0.00) | 0.56 (1.15)
  Cough, Week 78: number analyzed (Participants) | 2 | 7
  Cough, Week 78 | 0.25 (0.35) | 0.36 (1.03)
  Cough, Week 79: number analyzed (Participants) | 2 | 8
  Cough, Week 79 | 0.00 (0.00) | 0.63 (1.19)
  Cough, Week 80: number analyzed (Participants) | 2 | 9
  Cough, Week 80 | 0.25 (0.35) | 0.33 (0.90)
  Cough, Week 81: number analyzed (Participants) | 2 | 6
  Cough, Week 81 | 0.25 (0.35) | 0.58 (1.28)
  Cough, Week 82: number analyzed (Participants) | 1 | 6
  Cough, Week 82 | 0.00 | 0.25 (1.08)
  Cough, Week 83: number analyzed (Participants) | 1 | 6
  Cough, Week 83 | 0.00 | 0.67 (1.21)
  Cough, Week 84: number analyzed (Participants) | 1 | 7
  Cough, Week 84 | 0.50 | 0.29 (0.95)
  Cough, Week 85: number analyzed (Participants) | 1 | 8
  Cough, Week 85 | 0.00 | 0.38 (1.03)
  Cough, Week 86: number analyzed (Participants) | 1 | 7
  Cough, Week 86 | 0.00 | 0.57 (1.24)
  Cough, Week 87: number analyzed (Participants) | 1 | 7
  Cough, Week 87 | 0.00 | 0.64 (1.35)
  Cough, Week 88: number analyzed (Participants) | 0 | 7
  Cough, Week 88 |  | 0.64 (1.14)
  Cough, Week 89: number analyzed (Participants) | 0 | 5
  Cough, Week 89 |  | 0.50 (1.32)
  Cough, Week 90: number analyzed (Participants) | 0 | 7
  Cough, Week 90 |  | 0.43 (1.10)
  Cough, Week 91: number analyzed (Participants) | 0 | 7
  Cough, Week 91 |  | 0.50 (1.19)
  Cough, Week 92: number analyzed (Participants) | 0 | 6
  Cough, Week 92 |  | 0.67 (1.21)
  Cough, Week 93: number analyzed (Participants) | 0 | 7
  Cough, Week 93 |  | 0.79 (1.38)
  Cough, Week 94: number analyzed (Participants) | 0 | 5
  Cough, Week 94 |  | 0.30 (0.97)
  Cough, Week 95: number analyzed (Participants) | 0 | 6
  Cough, Week 95 |  | 0.67 (1.25)
  Cough, Week 96: number analyzed (Participants) | 0 | 6
  Cough, Week 96 |  | 0.58 (1.20)
  Cough, Week 97: number analyzed (Participants) | 0 | 7
  Cough, Week 97 |  | 0.57 (1.13)
  Cough, Week 98: number analyzed (Participants) | 0 | 6
  Cough, Week 98 |  | 0.67 (1.25)
  Cough, Week 99: number analyzed (Participants) | 0 | 4
  Cough, Week 99 |  | 0.25 (0.96)
  Cough, Week 100: number analyzed (Participants) | 0 | 5
  Cough, Week 100 |  | 0.60 (1.14)
  Cough, Week 101: number analyzed (Participants) | 0 | 6
  Cough, Week 101 |  | 0.50 (1.05)
  Cough, Week 102: number analyzed (Participants) | 0 | 5
  Cough, Week 102 |  | 0.50 (1.00)
  Cough, Week 103: number analyzed (Participants) | 0 | 4
  Cough, Week 103 |  | 0.25 (0.96)
  Cough, Week 104: number analyzed (Participants) | 0 | 3
  Cough, Week 104 |  | 0.00 (1.00)
  Cough, Week 105: number analyzed (Participants) | 0 | 3
  Cough, Week 105 |  | 0.33 (1.53)
  Cough, Week 106: number analyzed (Participants) | 0 | 2
  Cough, Week 106 |  | -0.50 (0.71)
  Cough, Week 107: number analyzed (Participants) | 0 | 3
  Cough, Week 107 |  | 0.00 (1.00)
  Cough, Week 108: number analyzed (Participants) | 0 | 2
  Cough, Week 108 |  | 0.00 (1.41)
  Cough, Week 109: number analyzed (Participants) | 0 | 2
  Cough, Week 109 |  | 0.50 (2.12)
  Cough, Week 110: number analyzed (Participants) | 0 | 2
  Cough, Week 110 |  | 0.50 (2.12)
  Cough, Week 111: number analyzed (Participants) | 0 | 2
  Cough, Week 111 |  | 0.50 (2.12)
  Cough, Week 112: number analyzed (Participants) | 0 | 2
  Cough, Week 112 |  | 0.00 (1.41)
  Cough, Week 113: number analyzed (Participants) | 0 | 2
  Cough, Week 113 |  | 0.50 (2.12)
  Cough, Week 114: number analyzed (Participants) | 0 | 2
  Cough, Week 114 |  | 0.50 (2.12)
  Cough, Week 115: number analyzed (Participants) | 0 | 2
  Cough, Week 115 |  | 0.50 (2.12)
  Cough, Week 116: number analyzed (Participants) | 0 | 2
  Cough, Week 116 |  | 0.50 (2.12)
  Cough, Week 117: number analyzed (Participants) | 0 | 2
  Cough, Week 117 |  | 0.50 (2.12)
  Cough, Week 118: number analyzed (Participants) | 0 | 2
  Cough, Week 118 |  | 0.50 (2.12)
  Cough, Week 119: number analyzed (Participants) | 0 | 2
  Cough, Week 119 |  | 0.50 (2.12)
  Cough, Week 120: number analyzed (Participants) | 0 | 1
  Cough, Week 120 |  | 2.00
  Cough, Week 121: number analyzed (Participants) | 0 | 1
  Cough, Week 121 |  | 2.00
  Cough, Week 122: number analyzed (Participants) | 0 | 1
  Cough, Week 122 |  | 2.00
  Cough, Week 123: number analyzed (Participants) | 0 | 1
  Cough, Week 123 |  | 2.00
  Cough, Week 124: number analyzed (Participants) | 0 | 1
  Cough, Week 124 |  | 2.00
  Cough, Week 125: number analyzed (Participants) | 0 | 1
  Cough, Week 125 |  | 2.00
  Cough, Week 126: number analyzed (Participants) | 0 | 1
  Cough, Week 126 |  | 2.00
  Cough, Week 127: number analyzed (Participants) | 0 | 1
  Cough, Week 127 |  | 2.00
  Cough, Week 128: number analyzed (Participants) | 0 | 1
  Cough, Week 128 |  | 2.00
  Cough, Week 129: number analyzed (Participants) | 0 | 1
  Cough, Week 129 |  | 2.00
  Cough, Week 130: number analyzed (Participants) | 0 | 1
  Cough, Week 130 |  | 2.00
  Cough, Week 131: number analyzed (Participants) | 0 | 1
  Cough, Week 131 |  | 2.00
  Dyspnoea, Week 1: number analyzed (Participants) | 44 | 47
  Dyspnoea, Week 1 | 0.42 (0.81) | 0.12 (0.76)
  Dyspnoea, Week 2: number analyzed (Participants) | 42 | 48
  Dyspnoea, Week 2 | 0.33 (0.73) | 0.29 (0.87)
  Dyspnoea, Week 3: number analyzed (Participants) | 44 | 49
  Dyspnoea, Week 3 | 0.25 (0.75) | 0.25 (0.97)
  Dyspnoea, Week 4: number analyzed (Participants) | 41 | 49
  Dyspnoea, Week 4 | 0.43 (0.87) | 0.28 (0.89)
  Dyspnoea, Week 5: number analyzed (Participants) | 39 | 47
  Dyspnoea, Week 5 | 0.55 (0.81) | 0.21 (1.00)
  Dyspnoea, Week 6: number analyzed (Participants) | 33 | 48
  Dyspnoea, Week 6 | 0.50 (0.68) | 0.21 (0.95)
  Dyspnoea, Week 7: number analyzed (Participants) | 30 | 44
  Dyspnoea, Week 7 | 0.63 (0.74) | 0.32 (1.08)
  Dyspnoea, Week 8: number analyzed (Participants) | 29 | 44
  Dyspnoea, Week 8 | 0.50 (0.64) | 0.25 (1.00)
  Dyspnoea, Week 9: number analyzed (Participants) | 31 | 47
  Dyspnoea, Week 9 | 0.46 (0.86) | 0.34 (1.01)
  Dyspnoea, Week 10: number analyzed (Participants) | 30 | 40
  Dyspnoea, Week 10 | 0.43 (0.80) | 0.49 (1.12)
  Dyspnoea, Week 11: number analyzed (Participants) | 29 | 34
  Dyspnoea, Week 11 | 0.36 (0.77) | 0.24 (0.97)
  Dyspnoea, Week 12: number analyzed (Participants) | 32 | 40
  Dyspnoea, Week 12 | 0.39 (0.82) | 0.35 (1.04)
  Dyspnoea, Week 13: number analyzed (Participants) | 28 | 38
  Dyspnoea, Week 13 | 0.43 (0.83) | 0.23 (0.94)
  Dyspnoea, Week 14: number analyzed (Participants) | 28 | 35
  Dyspnoea, Week 14 | 0.26 (0.88) | 0.26 (1.14)
  Dyspnoea, Week 15: number analyzed (Participants) | 30 | 40
  Dyspnoea, Week 15 | 0.36 (1.07) | 0.39 (1.22)
  Dyspnoea, Week 16: number analyzed (Participants) | 25 | 32
  Dyspnoea, Week 16 | 0.18 (0.82) | 0.26 (1.13)
  Dyspnoea, Week 17: number analyzed (Participants) | 27 | 34
  Dyspnoea, Week 17 | 0.48 (0.87) | 0.16 (1.17)
  Dyspnoea, Week 18: number analyzed (Participants) | 23 | 37
  Dyspnoea, Week 18 | 0.39 (0.65) | 0.21 (1.05)
  Dyspnoea, Week 19: number analyzed (Participants) | 22 | 32
  Dyspnoea, Week 19 | 0.29 (0.86) | 0.33 (1.12)
  Dyspnoea, Week 20: number analyzed (Participants) | 22 | 35
  Dyspnoea, Week 20 | 0.60 (0.87) | 0.23 (1.00)
  Dyspnoea, Week 21: number analyzed (Participants) | 18 | 36
  Dyspnoea, Week 21 | 0.27 (0.69) | 0.40 (0.93)
  Dyspnoea, Week 22: number analyzed (Participants) | 20 | 35
  Dyspnoea, Week 22 | 0.55 (0.92) | 0.22 (0.99)
  Dyspnoea, Week 23: number analyzed (Participants) | 16 | 33
  Dyspnoea, Week 23 | 0.34 (0.69) | 0.38 (0.98)
  Dyspnoea, Week 24: number analyzed (Participants) | 16 | 33
  Dyspnoea, Week 24 | 0.36 (1.02) | 0.42 (1.06)
  Dyspnoea, Week 25: number analyzed (Participants) | 11 | 29
  Dyspnoea, Week 25 | 0.22 (0.46) | 0.50 (1.14)
  Dyspnoea, Week 26: number analyzed (Participants) | 13 | 32
  Dyspnoea, Week 26 | 0.32 (0.82) | 0.28 (0.95)
  Dyspnoea, Week 27: number analyzed (Participants) | 11 | 32
  Dyspnoea, Week 27 | 0.35 (1.07) | 0.37 (1.04)
  Dyspnoea, Week 28: number analyzed (Participants) | 11 | 30
  Dyspnoea, Week 28 | 0.35 (0.92) | 0.45 (0.83)
  Dyspnoea, Week 29: number analyzed (Participants) | 12 | 28
  Dyspnoea, Week 29 | 0.20 (0.89) | 0.38 (0.85)
  Dyspnoea, Week 30: number analyzed (Participants) | 12 | 30
  Dyspnoea, Week 30 | 0.18 (0.96) | 0.54 (1.01)
  Dyspnoea, Week 31: number analyzed (Participants) | 11 | 29
  Dyspnoea, Week 31 | 0.18 (0.84) | 0.41 (0.86)
  Dyspnoea, Week 32: number analyzed (Participants) | 11 | 23
  Dyspnoea, Week 32 | 0.22 (1.00) | 0.58 (1.04)
  Dyspnoea, Week 33: number analyzed (Participants) | 13 | 26
  Dyspnoea, Week 33 | 0.20 (0.78) | 0.36 (0.96)
  Dyspnoea, Week 34: number analyzed (Participants) | 10 | 26
  Dyspnoea, Week 34 | 0.16 (0.79) | 0.28 (1.00)
  Dyspnoea, Week 35: number analyzed (Participants) | 11 | 27
  Dyspnoea, Week 35 | 0.11 (0.58) | 0.27 (1.02)
  Dyspnoea, Week 36: number analyzed (Participants) | 9 | 25
  Dyspnoea, Week 36 | 0.11 (0.86) | -0.02 (1.04)
  Dyspnoea, Week 37: number analyzed (Participants) | 8 | 23
  Dyspnoea, Week 37 | 0.28 (0.63) | 0.42 (1.13)
  Dyspnoea, Week 38: number analyzed (Participants) | 11 | 21
  Dyspnoea, Week 38 | 0.40 (0.76) | 0.50 (1.25)
  Dyspnoea, Week 39: number analyzed (Participants) | 9 | 22
  Dyspnoea, Week 39 | 0.27 (0.81) | 0.25 (0.86)
  Dyspnoea, Week 40: number analyzed (Participants) | 7 | 23
  Dyspnoea, Week 40 | 0.57 (0.76) | 0.44 (1.13)
  Dyspnoea, Week 41: number analyzed (Participants) | 7 | 20
  Dyspnoea, Week 41 | 0.31 (0.58) | 0.53 (1.17)
  Dyspnoea, Week 42: number analyzed (Participants) | 6 | 20
  Dyspnoea, Week 42 | 0.30 (0.55) | 0.52 (1.07)
  Dyspnoea, Week 43: number analyzed (Participants) | 5 | 20
  Dyspnoea, Week 43 | 0.40 (0.57) | 0.41 (1.18)
  Dyspnoea, Week 44: number analyzed (Participants) | 7 | 19
  Dyspnoea, Week 44 | 0.49 (0.60) | 0.31 (1.14)
  Dyspnoea, Week 45: number analyzed (Participants) | 4 | 21
  Dyspnoea, Week 45 | 0.65 (0.38) | 0.53 (1.04)
  Dyspnoea, Week 46: number analyzed (Participants) | 5 | 19
  Dyspnoea, Week 46 | 0.56 (0.71) | 0.37 (0.97)
  Dyspnoea, Week 47: number analyzed (Participants) | 4 | 18
  Dyspnoea, Week 47 | 0.30 (0.68) | 0.39 (0.92)
  Dyspnoea, Week 48: number analyzed (Participants) | 3 | 15
  Dyspnoea, Week 48 | 0.60 (0.72) | 0.39 (0.93)
  Dyspnoea, Week 49: number analyzed (Participants) | 3 | 17
  Dyspnoea, Week 49 | 1.40 (1.20) | 0.47 (0.76)
  Dyspnoea, Week 50: number analyzed (Participants) | 5 | 15
  Dyspnoea, Week 50 | 0.24 (0.59) | 0.53 (0.96)
  Dyspnoea, Week 51: number analyzed (Participants) | 4 | 16
  Dyspnoea, Week 51 | 1.05 (1.02) | 0.59 (1.02)
  Dyspnoea, Week 52: number analyzed (Participants) | 4 | 13
  Dyspnoea, Week 52 | 1.10 (1.01) | 0.72 (1.20)
  Dyspnoea, Week 53: number analyzed (Participants) | 5 | 12
  Dyspnoea, Week 53 | 0.76 (1.28) | 0.40 (1.01)
  Dyspnoea, Week 54: number analyzed (Participants) | 4 | 14
  Dyspnoea, Week 54 | 1.10 (1.16) | 0.63 (1.02)
  Dyspnoea, Week 55: number analyzed (Participants) | 3 | 13
  Dyspnoea, Week 55 | 1.00 (0.53) | 0.72 (1.13)
  Dyspnoea, Week 56: number analyzed (Participants) | 4 | 14
  Dyspnoea, Week 56 | 0.40 (0.86) | 0.61 (1.07)
  Dyspnoea, Week 57: number analyzed (Participants) | 3 | 13
  Dyspnoea, Week 57 | 0.53 (0.61) | 0.45 (1.02)
  Dyspnoea, Week 58: number analyzed (Participants) | 3 | 13
  Dyspnoea, Week 58 | 0.80 (0.53) | 0.60 (1.20)
  Dyspnoea, Week 59: number analyzed (Participants) | 3 | 9
  Dyspnoea, Week 59 | 0.60 (0.72) | 0.18 (1.08)
  Dyspnoea, Week 60: number analyzed (Participants) | 2 | 13
  Dyspnoea, Week 60 | 1.20 (1.13) | 0.57 (0.89)
  Dyspnoea, Week 61: number analyzed (Participants) | 3 | 14
  Dyspnoea, Week 61 | 0.73 (0.76) | 0.54 (1.00)
  Dyspnoea, Week 62: number analyzed (Participants) | 3 | 14
  Dyspnoea, Week 62 | 0.67 (0.83) | 0.66 (1.11)
  Dyspnoea, Week 63: number analyzed (Participants) | 2 | 12
  Dyspnoea, Week 63 | 0.30 (0.42) | 0.77 (0.80)
  Dyspnoea, Week 64: number analyzed (Participants) | 1 | 10
  Dyspnoea, Week 64 | 0.20 | 0.66 (1.07)
  Dyspnoea, Week 65: number analyzed (Participants) | 1 | 13
  Dyspnoea, Week 65 | 0.60 | 0.94 (1.28)
  Dyspnoea, Week 66: number analyzed (Participants) | 1 | 11
  Dyspnoea, Week 66 | 0.40 | 0.67 (1.31)
  Dyspnoea, Week 67: number analyzed (Participants) | 2 | 11
  Dyspnoea, Week 67 | 0.50 (0.14) | 0.33 (0.87)
  Dyspnoea, Week 68: number analyzed (Participants) | 2 | 9
  Dyspnoea, Week 68 | 0.20 (0.28) | 0.82 (1.56)
  Dyspnoea, Week 69: number analyzed (Participants) | 2 | 10
  Dyspnoea, Week 69 | 0.30 (0.42) | 0.74 (1.11)
  Dyspnoea, Week 70: number analyzed (Participants) | 2 | 11
  Dyspnoea, Week 70 | 0.30 (0.42) | 0.75 (1.16)
  Dyspnoea, Week 71: number analyzed (Participants) | 2 | 10
  Dyspnoea, Week 71 | 0.10 (0.14) | 0.84 (1.19)
  Dyspnoea, Week 72: number analyzed (Participants) | 1 | 12
  Dyspnoea, Week 72 | 0.00 | 0.80 (1.09)
  Dyspnoea, Week 73: number analyzed (Participants) | 1 | 11
  Dyspnoea, Week 73 | 0.00 | 0.67 (1.11)
  Dyspnoea, Week 74: number analyzed (Participants) | 2 | 9
  Dyspnoea, Week 74 | 0.20 (0.28) | 0.89 (1.35)
  Dyspnoea, Week 75: number analyzed (Participants) | 2 | 9
  Dyspnoea, Week 75 | 0.30 (0.42) | 0.71 (1.31)
  Dyspnoea, Week 76: number analyzed (Participants) | 1 | 8
  Dyspnoea, Week 76 | 0.30 (0.42) | 0.53 (1.05)
  Dyspnoea, Week 77: number analyzed (Participants) | 2 | 8
  Dyspnoea, Week 77 | 0.40 (0.57) | 0.65 (1.55)
  Dyspnoea, Week 78: number analyzed (Participants) | 2 | 7
  Dyspnoea, Week 78 | 0.30 (0.14) | 0.40 (1.11)
  Dyspnoea, Week 79: number analyzed (Participants) | 2 | 8
  Dyspnoea, Week 79 | 0.10 (0.14) | 0.55 (1.25)
  Dyspnoea, Week 80: number analyzed (Participants) | 2 | 9
  Dyspnoea, Week 80 | 0.50 (0.71) | 0.69 (1.43)
  Dyspnoea, Week 81: number analyzed (Participants) | 2 | 6
  Dyspnoea, Week 81 | 0.40 (0.57) | 0.53 (1.53)
  Dyspnoea, Week 82: number analyzed (Participants) | 1 | 6
  Dyspnoea, Week 82 | 0.60 | 0.53 (1.09)
  Dyspnoea, Week 83: number analyzed (Participants) | 1 | 6
  Dyspnoea, Week 83 | 0.60 | 0.87 (1.28)
  Dyspnoea, Week 84: number analyzed (Participants) | 1 | 7
  Dyspnoea, Week 84 | 0.80 | 0.89 (1.13)
  Dyspnoea, Week 85: number analyzed (Participants) | 1 | 8
  Dyspnoea, Week 85 | 0.60 | 0.83 (1.27)
  Dyspnoea, Week 86: number analyzed (Participants) | 1 | 7
  Dyspnoea, Week 86 | 0.40 | 0.66 (1.33)
  Dyspnoea, Week 87: number analyzed (Participants) | 1 | 7
  Dyspnoea, Week 87 | 0.40 | 0.66 (1.23)
  Dyspnoea, Week 88: number analyzed (Participants) | 0 | 7
  Dyspnoea, Week 88 |  | 1.20 (1.43)
  Dyspnoea, Week 89: number analyzed (Participants) | 0 | 5
  Dyspnoea, Week 89 |  | 0.56 (1.05)
  Dyspnoea, Week 90: number analyzed (Participants) | 0 | 7
  Dyspnoea, Week 90 |  | 0.74 (1.38)
  Dyspnoea, Week 91: number analyzed (Participants) | 0 | 7
  Dyspnoea, Week 91 |  | 0.51 (1.00)
  Dyspnoea, Week 92: number analyzed (Participants) | 0 | 6
  Dyspnoea, Week 92 |  | 0.87 (1.26)
  Dyspnoea, Week 93: number analyzed (Participants) | 0 | 7
  Dyspnoea, Week 93 |  | 1.20 (1.39)
  Dyspnoea, Week 94: number analyzed (Participants) | 0 | 5
  Dyspnoea, Week 94 |  | 0.48 (0.99)
  Dyspnoea, Week 95: number analyzed (Participants) | 0 | 6
  Dyspnoea, Week 95 |  | 0.87 (1.32)
  Dyspnoea, Week 96: number analyzed (Participants) | 0 | 6
  Dyspnoea, Week 96 |  | 1.13 (1.24)
  Dyspnoea, Week 97: number analyzed (Participants) | 0 | 7
  Dyspnoea, Week 97 |  | 1.26 (1.35)
  Dyspnoea, Week 98: number analyzed (Participants) | 0 | 6
  Dyspnoea, Week 98 |  | 0.80 (1.19)
  Dyspnoea, Week 99: number analyzed (Participants) | 0 | 4
  Dyspnoea, Week 99 |  | 0.70 (1.58)
  Dyspnoea, Week 100: number analyzed (Participants) | 0 | 5
  Dyspnoea, Week 100 |  | 0.88 (1.38)
  Dyspnoea, Week 101: number analyzed (Participants) | 0 | 6
  Dyspnoea, Week 101 |  | 1.13 (1.54)
  Dyspnoea, Week 102: number analyzed (Participants) | 0 | 5
  Dyspnoea, Week 102 |  | 0.96 (1.58)
  Dyspnoea, Week 103: number analyzed (Participants) | 0 | 4
  Dyspnoea, Week 103 |  | 0.55 (1.68)
  Dyspnoea, Week 104: number analyzed (Participants) | 0 | 3
  Dyspnoea, Week 104 |  | 1.07 (1.33)
  Dyspnoea, Week 105: number analyzed (Participants) | 0 | 3
  Dyspnoea, Week 105 |  | 1.07 (1.33)
  Dyspnoea, Week 106: number analyzed (Participants) | 0 | 2
  Dyspnoea, Week 106 |  | 0.40 (0.28)
  Dyspnoea, Week 107: number analyzed (Participants) | 0 | 3
  Dyspnoea, Week 107 |  | 1.13 (1.63)
  Dyspnoea, Week 108: number analyzed (Participants) | 0 | 2
  Dyspnoea, Week 108 |  | 1.50 (1.56)
  Dyspnoea, Week 109: number analyzed (Participants) | 0 | 2
  Dyspnoea, Week 109 |  | 1.30 (1.27)
  Dyspnoea, Week 110: number analyzed (Participants) | 0 | 2
  Dyspnoea, Week 110 |  | 1.50 (1.56)
  Dyspnoea, Week 111: number analyzed (Participants) | 0 | 2
  Dyspnoea, Week 111 |  | 1.60 (1.41)
  Dyspnoea, Week 112: number analyzed (Participants) | 0 | 2
  Dyspnoea, Week 112 |  | 1.50 (1.56)
  Dyspnoea, Week 113: number analyzed (Participants) | 0 | 2
  Dyspnoea, Week 113 |  | 1.50 (1.56)
  Dyspnoea, Week 114: number analyzed (Participants) | 0 | 2
  Dyspnoea, Week 114 |  | 1.60 (1.70)
  Dyspnoea, Week 115: number analyzed (Participants) | 0 | 2
  Dyspnoea, Week 115 |  | 1.40 (1.41)
  Dyspnoea, Week 116: number analyzed (Participants) | 0 | 2
  Dyspnoea, Week 116 |  | 1.30 (1.27)
  Dyspnoea, Week 117: number analyzed (Participants) | 0 | 2
  Dyspnoea, Week 117 |  | 1.50 (1.56)
  Dyspnoea, Week 118: number analyzed (Participants) | 0 | 2
  Dyspnoea, Week 118 |  | 1.30 (1.27)
  Dyspnoea, Week 119: number analyzed (Participants) | 0 | 2
  Dyspnoea, Week 119 |  | 1.50 (1.56)
  Dyspnoea, Week 120: number analyzed (Participants) | 0 | 1
  Dyspnoea, Week 120 |  | 2.20
  Dyspnoea, Week 121: number analyzed (Participants) | 0 | 1
  Dyspnoea, Week 121 |  | 2.40
  Dyspnoea, Week 122: number analyzed (Participants) | 0 | 1
  Dyspnoea, Week 122 |  | 2.20
  Dyspnoea, Week 123: number analyzed (Participants) | 0 | 1
  Dyspnoea, Week 123 |  | 2.20
  Dyspnoea, Week 124: number analyzed (Participants) | 0 | 1
  Dyspnoea, Week 124 |  | 2.20
  Dyspnoea, Week 125: number analyzed (Participants) | 0 | 1
  Dyspnoea, Week 125 |  | 2.20
  Dyspnoea, Week 126: number analyzed (Participants) | 0 | 1
  Dyspnoea, Week 126 |  | 2.20
  Dyspnoea, Week 127: number analyzed (Participants) | 0 | 1
  Dyspnoea, Week 127 |  | 2.20
  Dyspnoea, Week 128: number analyzed (Participants) | 0 | 1
  Dyspnoea, Week 128 |  | 2.20
  Dyspnoea, Week 129: number analyzed (Participants) | 0 | 1
  Dyspnoea, Week 129 |  | 2.20
  Dyspnoea, Week 130: number analyzed (Participants) | 0 | 1
  Dyspnoea, Week 130 |  | 2.20
  Dyspnoea, Week 131: number analyzed (Participants) | 0 | 1
  Dyspnoea, Week 131 |  | 2.20

15. Secondary Outcome: TTD as Assessed Using EORTC QLQ Supplementary Lung Cancer Module (EORTC QLQ-LC13) in the TC3 or IC3-WT Populations
Description: TTD in patient-reported lung cancer symptoms, defined as time from randomization to deterioration (10-point change) in any of the following symptom subscales (cough, dyspnea [multi-item scale], and chest pain), whichever occurs first, as measured by the EORTC QLQ-LC13. EORTC QLQ-LC13 module incorporates one multi-item scale to assess dyspnea and a series of single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis.
Time Frame: Baseline until data cut-off on 10 September 2018 (up to approximately 38 months)
Population: Analysis was performed for the TC3 or IC3-WT Populations.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 98 | 107
Months
  Cough | NA [NA to NA] — Median TTD is not estimable by Kaplan-Meier method due to insufficient observed events. Lower/Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events | NA [21.5 to NA] — Median TTD is not estimable by Kaplan-Meier method due to insufficient number of observed events. Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events.
  Dyspnea | 11.8 [6.8 to 19.5] | 11.1 [7.0 to NA] — Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events.
  Chest pain | NA [NA to NA] — Median TTD is not estimable by Kaplan-Meier method due to insufficient number of observed events. Lower/Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events. | NA [NA to NA] — Median TTD is not estimable by Kaplan-Meier method due to insufficient number of observed events. Lower/Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events.
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; Cough for TC3 or IC3-WT Populations; Test type: Superiority — Stratified analysis; Hazard Ratio (HR) = 0.984, 95% CI 2-sided [0.477 to 2.030]
Statistical Analysis 2: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; Dyspnea for TC3 or IC3-WT Populations; Test type: Superiority — Stratified analysis; Hazard Ratio (HR) = 0.955, 95% CI 2-sided [0.569 to 1.604]
Statistical Analysis 3: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; Chest pain for TC3 or IC3-WT Populations; Test type: Superiority — Stratified analysis; Hazard Ratio (HR) = 1.024, 95% CI 2-sided [0.472 to 2.222]

16. Secondary Outcome: OS in Participants With PD-L1 Expression
Description: OS is defined as the time from randomization to death from any cause.
Time Frame: From randomization to death from any cause until data cut-off on 10 September 2018 (up to approximately 38 months)
Population: Analysis was performed for participants with PD-L1 Expression of PD-L1 status by SP263 >=50%, SP263 >=25%, SP263 >=1% in the Intent-to-Treat Wild Type Population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 210 | 212
Months
  SP263 >=50%-WT Population: number analyzed (Participants) | 143 | 150
  SP263 >=50%-WT Population | 16.1 [9.8 to 17.4] | 19.5 [13.8 to NA] — Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events.
  SP263 >=25%-WT Population: number analyzed (Participants) | 168 | 168
  SP263 >=25%-WT Population | 12.6 [9.1 to 17.0] | 18.2 [13.3 to NA] — Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events.
  SP263 =1%-WT Population | 14.0 [9.8 to 16.5] | 17.8 [12.8 to 23.1]
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; SP263 >=50%-WT Population; Test type: Superiority — Unstratified analysis; Hazard Ratio (HR) = 0.707, 95% CI 2-sided [0.500 to 1.000]
Statistical Analysis 2: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; SP263 >=25%-WT Population; Test type: Superiority — Unstratified analysis; Hazard Ratio (HR) = 0.693, 95% CI 2-sided [0.502 to 0.956]
Statistical Analysis 3: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; SP263 >=1%-WT Population; Test type: Superiority — Unstratified analysis; Hazard Ratio (HR) = 0.768, 95% CI 2-sided [0.579 to 1.018]

17. Secondary Outcome: Investigator-Assessed PFS in Participants With PD-L1 Expression According to RECIST v1.1
Description: Investigator-assessed PFS according to RECIST v1.1 in the PD-L1 (defined with SP263 IHC assay)
Time Frame: as for outcome 3
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 210 | 212
Months
  SP263 >=50%-WT Population: number analyzed (Participants) | 143 | 150
  SP263 >=50%-WT Population | 4.9 [4.0 to 5.6] | 7.0 [5.6 to 8.7]
  SP263 >=25%-WT Population: number analyzed (Participants) | 168 | 168
  SP263 >=25%-WT Population | 4.9 [4.2 to 5.6] | 6.9 [5.6 to 8.4]
  SP263 >=1%-WT Population | 5.4 [4.4 to 5.7] | 6.8 [5.5 to 8.0]
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; SP263 >=50%-WT Population; Test type: Superiority — Unstratified analysis; Hazard Ratio (HR) = 0.674, 95% CI 2-sided [0.511 to 0.890]
Statistical Analysis 2: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; SP263 >=25%-WT Population; Test type: Superiority — Unstratified analysis; Hazard Ratio (HR) = 0.698, 95% CI 2-sided [0.539 to 0.904]
Statistical Analysis 3: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; SP263 >=1%-WT Population; Test type: Superiority — Unstratified analysis; Hazard Ratio (HR) = 0.725, 95% CI 2-sided [0.577 to 0.910]

18. Secondary Outcome: OS in Participants With Blood Tumor Mutational Burden (bTMB)
Description: OS is defined as the time from randomization to death from any cause.
Time Frame: From randomization to death from any cause until data cut-off on 10 September 2018 (up to approximately 38 months)
Population: Analysis was performed for the bTMB subpopulations in the Intent-to-Treat Wild Type population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 83 | 92
Months
  bTMB >=10-WT Population | 10.3 [7.1 to 16.9] | 11.2 [7.9 to NA] — Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events.
  bTMB >=16-WT Population: number analyzed (Participants) | 45 | 42
  bTMB >=16-WT Population | 8.5 [5.8 to NA] — Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events. | 13.9 [10.8 to NA] — Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events.
  bTMB >=20-WT Population: number analyzed (Participants) | 29 | 27
  bTMB >=20-WT Population | 10.5 [5.8 to NA] — Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events. | 17.2 [10.8 to NA] — Upper limit of 95% confidence interval is not estimable by Brookmeyer and Crowley method due to insufficient number of observed events.
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; bTMB >=10-WT Population; Test type: Superiority — Unstratified analysis; Hazard Ratio (HR) = 0.867, 95% CI 2-sided [0.578 to 1.301]
Statistical Analysis 2: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; bTMB >=16-WT Population; Test type: Superiority — Unstratified analysis; Hazard Ratio (HR) = 0.748, 95% CI 2-sided [0.414 to 1.351]
Statistical Analysis 3: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; bTMB >=20-WT Population; Test type: Superiority — Unstratified analysis; Hazard Ratio (HR) = 0.770, 95% CI 2-sided [0.362 to 1.638]

19. Secondary Outcome: Investigator-Assessed PFS in Participants With bTMB According to RECIST v1.1
Description: PFS according to RECIST v1.1 in the bTMB subpopulations.
Time Frame: as for outcome 3
Population: Analysis was performed for participants with bTMB >=10 Intent-to-treat Wild Type Population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 83 | 92
Months
  bTMB >=10-WT Population | 4.3 [3.1 to 5.4] | 5.5 [2.8 to 6.8]
  bTMB >=16-WT Population: number analyzed (Participants) | 45 | 42
  bTMB >=16-WT Population | 4.4 [2.8 to 5.7] | 6.8 [4.3 to 11.6]
  bTMB >=20-WT Population: number analyzed (Participants) | 29 | 27
  bTMB >=20-WT Population | 5.2 [3.2 to 6.4] | 6.8 [4.3 to 17.2]
Statistical Analysis 1: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; bTMB >=10-WT Population; Test type: Superiority — Unstratified analysis; Hazard Ratio (HR) = 0.743, 95% CI 2-sided [0.525 to 1.052]
Statistical Analysis 2: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; bTMB >=16-WT Population; Test type: Superiority — Unstratified analysis; Hazard Ratio (HR) = 0.553, 95% CI 2-sided [0.331 to 0.924]
Statistical Analysis 3: Comparison: Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) vs Atezolizumab; bTMB >=20-WT Population; Test type: Superiority — Unstratified analysis; Hazard Ratio (HR) = 0.560, 95% CI 2-sided [0.295 to 1.062]

20. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Atezolizumab
Time Frame: Prior to infusion (0 hour) on Day 1 of Cycles 2, 3, 4, 8, 16, and every eighth cycle thereafter, and at treatment discontinuation until data cut-off on 10 September 2018 (up to approximately 38 months) (cycle duration = 21 days)
Population: PK analyses was based on PK observations from all randomized participants who received atezolizumab and provided at least one PK sample that was evaluable.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (μg/ mL)
Arm/Group | Atezolizumab
Number analyzed (Participants) | 256
micrograms per milliliter (μg/ mL)
  Cycle 2 Day 1 | 76.7 (57.6)
  Cycle 3 Day 1: number analyzed (Participants) | 215
  Cycle 3 Day 1 | 121 (57.7)
  Cycle 4 Day 1: number analyzed (Participants) | 207
  Cycle 4 Day 1 | 154 (90.1)
  Cycle 8 Day 1: number analyzed (Participants) | 145
  Cycle 8 Day 1 | 201 (98.6)
  Cycle 16 Day 1: number analyzed (Participants) | 67
  Cycle 16 Day 1 | 213 (102)
  Cycle 24 Day 1: number analyzed (Participants) | 31
  Cycle 24 Day 1 | 245 (128)
  Cycle 32 Day 1: number analyzed (Participants) | 10
  Cycle 32 Day 1 | 276 (110)
  Cycle 40 Day 1: number analyzed (Participants) | 5
  Cycle 40 Day 1 | 252 (160)
  Cycle 48 Day 1: number analyzed (Participants) | 1
  Cycle 48 Day 1 | 555 (NA) — Not estimable because there is only 1 participant.
  Treatment Discontinuation Visit: number analyzed (Participants) | 100
  Treatment Discontinuation Visit | 121 (88.8)

21. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Atezolizumab
Time Frame: 0 hour (predose) and 30 minutes after atezolizumab infusion on Day 1 (infusion duration = up to 1 hour)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (μg/ mL)
Arm/Group | Atezolizumab
Number analyzed (Participants) | 270
micrograms per milliliter (μg/ mL) | 411 (163)

22. Secondary Outcome: Percentage of Participants With at Least One Adverse Event
Description: Percentage of participants with at least one adverse event.
Time Frame: Baseline up to until data cut-off on 8 March 2022 (up to approximately 79.5 months)
Population: Safety analyses included treated participants, defined as randomized participants who received any amount of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
Number analyzed (Participants) | 263 | 286
Percentage of participants | 95.1 | 92.3

23. Secondary Outcome: Percentage of Participants With Anti-therapeutic Antibodies (ATAs)
Time Frame: Baseline until data cut-off on 10 September 2018 (up to approximately 38 months)
Population: The baseline ADA-evaluable population included participants who had a baseline ADA result and had received at least one dose of atezolizumab. The post-baseline ADA evaluable population included participants who had at least one post-baseline ADA result and had received at least one dose of atezolizumab.
Measure: Number; unit: Percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 282
Percentage of participants
  Baseline evaluable participants | 1.4
  Post-baseline evaluable participants: number analyzed (Participants) | 267
  Post-baseline evaluable participants | 24.3

ADVERSE EVENTS:
Time Frame: From the first study drug until the data cut-off on 8 March 2022 (up to approximately 79.5 months)
Description: All-cause mortality reported for deaths that occurred during study based on ITT, which included all randomized participants. Serious & other adverse events reported based on safety population, which included participants who received any amount of any study drug.
Arm/Group | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 211/287 | 201/285
Serious Adverse Events (participants affected / at risk) | 77/263 | 97/286
Other Adverse Events (participants affected / at risk) | 230/263 | 238/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) (N=263) | Atezolizumab (N=286)
Anaemia (Blood and lymphatic system disorders) | 10 (15) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (10) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (2)
Autoimmune myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Glucocorticoid deficiency (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 4 (5)
Swelling (General disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (2)
Immune system disorder (Immune system disorders) | 0 (0) | 1 (2)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 1 (2)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (3)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Muscle abscess (Infections and infestations) | 1 (1) | 0 (0)
Mycotic endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 14 (14) | 15 (25)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 4 (5) | 3 (3)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 1 (2) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Thrombosis in device (Product Issues) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Ketonuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (10)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Autoimmune dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bacterial colitis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 1 (1)
Langerhans' cell histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Vein disorder (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (Carboplatin/ Cisplatin) + (Pemetrexed/ Gemcitabine) (N=263) | Atezolizumab (N=286)
Anaemia (Blood and lymphatic system disorders) | 120 (153) | 50 (73)
Leukopenia (Blood and lymphatic system disorders) | 21 (31) | 4 (6)
Neutropenia (Blood and lymphatic system disorders) | 71 (128) | 5 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 40 (62) | 8 (8)
Hypothyroidism (Endocrine disorders) | 3 (3) | 27 (28)
Constipation (Gastrointestinal disorders) | 58 (75) | 42 (48)
Diarrhoea (Gastrointestinal disorders) | 30 (39) | 39 (55)
Nausea (Gastrointestinal disorders) | 88 (148) | 42 (49)
Stomatitis (Gastrointestinal disorders) | 14 (16) | 12 (14)
Vomiting (Gastrointestinal disorders) | 34 (45) | 21 (27)
Asthenia (General disorders) | 47 (66) | 41 (58)
Chest pain (General disorders) | 10 (10) | 21 (28)
Fatigue (General disorders) | 47 (57) | 44 (47)
Pyrexia (General disorders) | 25 (30) | 40 (58)
Nasopharyngitis (Infections and infestations) | 7 (8) | 22 (37)
Alanine aminotransferase increased (Investigations) | 16 (17) | 30 (34)
Aspartate aminotransferase increased (Investigations) | 11 (12) | 29 (35)
Blood creatinine increased (Investigations) | 27 (33) | 9 (12)
Neutrophil count decreased (Investigations) | 19 (27) | 0 (0)
Platelet count decreased (Investigations) | 21 (30) | 1 (1)
Weight decreased (Investigations) | 15 (15) | 25 (27)
White blood cell count decreased (Investigations) | 14 (24) | 3 (17)
Decreased appetite (Metabolism and nutrition disorders) | 50 (61) | 50 (65)
Hyponatraemia (Metabolism and nutrition disorders) | 12 (19) | 19 (29)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 31 (46)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (15) | 26 (28)
Headache (Nervous system disorders) | 18 (20) | 31 (32)
Insomnia (Psychiatric disorders) | 15 (16) | 22 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (27) | 36 (48)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 (32) | 41 (48)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 23 (25)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (16) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 25 (33)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 23 (26)
Oedema peripheral (General disorders) | 16 (18) | 13 (14)
Hyperglycaemia (Metabolism and nutrition disorders) | 15 (17) | 12 (18)
Dizziness (Nervous system disorders) | 14 (18) | 9 (9)
Pneumonia (Infections and infestations) | 8 (8) | 15 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-02-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT02409342/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT02409342/SAP_001.pdf